# **Cover Page for Statistical Analysis Plan**

| Sponsor name: | Novo Nordisk A/S |
|---|---|
| NCT number | NCT05064735 |
| Sponsor trial ID: | NN9536-4578 |
| Official title of study: | Effect of subcutaneous semaglutide 2.4 mg once-weekly compared to placebo in subjects with obesity and knee osteoarthritis |
| Document date* | 13 November 2023 |

\*Document date refers to the date on which the document was most recently updated.

Note: The date in the header of Page 2 is the date of compilation of the documents and not of an update to content.

| Semaglutide s.c. 2.4 mg once weekly |
|-------------------------------------|
| Study ID: NN9536-4578 (Knee OA) |
| Clinical Study Report |
| Appendix 9.1.9 |


Date: Version: Status: 12 January 2024 Novo Nordisk 1.0 Final

## 9.1.9 Documentation of statistical methods

# List of contents

| Statistical analysis plan | Link |
|--------------------------------------------------|------|
| Memo on Post-hoc analysis for responder endpoint | Link |
| MedDRA searches | Link |
| Psychometric Analysis Plan | Link |

Redacted statistical analysis plan includes redaction of personal identifiable and company confidential information.

Statistical Analysis Plan Trial ID: NN9536-4578


 Date:
 13 November 2023
 Novo Nordisk

 Version:
 6.0

 Status:
 Final

 Page:
 1 of 28

## Statistical Analysis Plan

**Trial ID: NN9536-4578** 

Effect of subcutaneous semaglutide 2.4 mg once-weekly compared to placebo in subjects with obesity and knee osteoarthritis

Author

**Biostatistics** 

This confidential document is the property of Novo Nordisk. No unpublished information contained herein may be disclosed without prior written approval from Novo Nordisk. Access to this document must be restricted to relevant parties.

SAP NN9536-4578 SAP 1 of 28

Statistical Analysis Plan Trial ID: NN9536-4578


Date: Version: Status: Page:

13 November 2023 Novo Nordisk 6.0

6.0 Final 2 of 28

# Table of contents Page

| Γ | able of | f contents | S | | 2 |
|---|---|---|---|---|---|
| Li | ist of a | ıbbreviat | ions | | 3 |
| V | ersion | history | ••••• | | 4 |
| 1 | | • | | | |
| | 1.1 | | | | |
| | | 1.1.1 | Objective | (s) | 8 |
| | | | 1.1.1.1 | Primary objective | 8 |
| | | | 1.1.1.2 | Secondary objectives | 8 |
| | | | 1.1.1.3 | Exploratory objectives | 8 |
| | | 1.1.2 | Estimands | s | 8 |
| | | | 1.1.2.1 | Primary estimand | |
| | | | 1.1.2.2 | Additional estimand | |
| | | 1.1.3 | Endpoints | S | |
| | | | 1.1.3.1 | Primary endpoints | |
| | | | 1.1.3.2 | Confirmatory secondary endpoints | |
| | | | 1.1.3.3 | Supportive secondary endpoints | |
| | | | 1.1.3.4 | Exploratory endpoint(s) | |
| | | 1.1.4 | | rial | |
| | 1.2 | Scope of | f the statisti | ical analysis plan | 12 |
| 2 | Stati | stical con | siderations | S | 13 |
| | 2.1 | | | es | |
| | 2.2 | | | ination | |
| | 2.3 | Definition | on of analys | sis sets | 16 |
| | 2.4 | Statistic | | | |
| | | 2.4.1 | General c | onsiderations | 17 |
| | | 2.4.2 | Primary e | ndpoint(s) | 18 |
| | | 2.4.3 | | y endpoints | 22 |
| | | | 2.4.3.1 | Confirmatory secondary endpoints | |
| | | | 2.4.3.2 | Supportive secondary endpoints | |
| | | 2.4.4 | Explorato | ry endpoints | 26 |
| 2 | Dofo | nonaoc | | | 10 |

Statistical Analysis Plan

Trial ID: NN9536-4578

Date: 13 November 2023 | Novo Nordisk
Version: 6.0

| CONFIDENTIAL | Version: 6.0 | Status: Final |

### List of abbreviations

AE adverse event

ANCOVA analysis of covariance
BMI body mass index
FAS full analysis set

ICH International Council for Harmonisation

J2R-MI jump to reference multiple imputation

*LAO-OT* last available observation during the on-treatment period

MedDRAMedical Dictionary for Regulatory ActivitiesMMRMmixed model for repeated measurements

NRS numerical rating scale

NSAIDs non-steroidal anti-inflammatory drugs

OA osteoarthritis OR odds ratio

PYE patient years of exposure
PYO patient years of observation

RD-MI retrieved dropout multiple imputation

SAE serious adverse event
SAP statistical analysis plan
SAS safety analysis set
SD standard deviation

SF-36 Short Form (36) Health Survey
TEAE treatment-emergent adverse event
TP-MI tipping-point multiple imputation

VAS visual analogue scale

WOMAC Western Ontario McMasters Osteoarthritis Index

SAP NN9536-4578 SAP 3 of 28

Statistical Analysis Plan
Trial ID: NN9536-4578

Date: 13 November 2023 Version: 6.0 Status: Final 

# **Version history**

This statistical analysis plan (SAP) is based on the updated protocol for trial NN9536-4578 "Effect of subcutaneous semaglutide 2.4 mg once-weekly compared to placebo in subjects with obesity and knee osteoarthritis", version 3.0 (21 April 2021).

| SAP version | Change | Rationale |
|---|---|---|
| 1.0<br>(03 August<br>2020) | Not applicable | Original version |
| 2.0<br>(03 May 2021) | The following supportive secondary endpoints have been added: • Amount of allowed rescue analgesics used during wash out • Change in pain intensity (NRS) • Achieving WOMAC pain reduction ≥30% (yes/no) • Achieving WOMAC pain reduction ≥50% (yes/no) • Achieving pain intensity (NRS) reduction ≥30% (yes/no) • Achieving pain intensity (NRS) reduction ≥50% (yes/no) The following supportive secondary endpoints are no longer in scope: • Change in body weight from baseline to week 28 • Change in WOMAC pain score from baseline to week 28 The exploratory endpoint "Change in pain medication (decrease/no change/increase)" has been renamed to "Change in pain medication" with dose as units. The following supportive secondary endpoints have been recategorized as exploratory endpoints: • Change in SF-36 role-physical score • Change in SF-36 social functioning score • Change in SF-36 social functioning score • Change in SF-36 mental health score | The overall rationale for preparing protocol version 3.0 was to include a pain and pain medication diary, to update supportive secondary endpoints and adjust WOMAC assessments with respect to frequency and recall period. |
| 3.0<br>(20 September<br>2021) | It has been specified in section 2.4.1 how the composite WOMAC scores are derived. It has been specified in more detail how missing WOMAC pain scores are handled in section 2.4.2 and 2.4.3.2, 2.4.3. For the endpoints related to change in WOMAC scores it is specified that imputation of missing values is done at the item level and not at the composite score level. | Correspondence with<br>the Food and Drug<br>Administration, US,<br>has prompted further<br>specification of how<br>missing data in the<br>WOMAC |

SAP NN9536-4578 SAP 4 of 28

Statistical Analysis Plan Trial ID: NN9536-4578

EudraCT No: 2017-003436-36


Date: Version: Status: Page: 13 November 2023 | **Novo Nordisk** 6.0

6.0 Final 5 of 28

| | · | , |
|---|---|---|
| | For the tipping-point multiple imputation analysis of the WOMAC pain score, the penalties added has been changed from -50/50 to -5/5 since WOMAC scores will be reported on a 0-10 point scale and not on a 0-100 point scale. In section 2.2 the following sentence has been deleted: "It is planned that the WOMAC scores (derived from NRS responses) will be transformed to a 0-100 range based on which the corresponding endpoints will be calculated." | questionnaire are handled. |
| 4.0<br>(28 February<br>2022) | The final reporting scale of WOMAC scores was set to be on the 0-100 range in order to comply with the protocol, specifically the randomisation criterion:" A score of at least 40 on the WOMAC version 3.1 pain subscale (range 0-100 normalised Numerical Rating Scale (NRS))". In consequence • the following sentence was again added to section 2.2: "It is planned that the WOMAC scores (derived from NRS responses) will be transformed to a 0-100 range based on which the corresponding endpoints will be calculated.", • section 2.4.1 describing how the composite WOMAC scores are derived was updated to reflect final reporting scale, i.e. normalisation to 0-100, • for the tipping-point multiple imputation analysis of the WOMAC pain score, the penalties were changed back from -5/5 to -50/50 since WOMAC scores will be reported on a 0-100 point scale. The following endpoints were added to section 1.1.3.3: "Subject achieving threshold(s) for clinically meaningful within-subject change in WOMAC pain score" (similar for WOMAC physical function score and SF-36 physical functioning score), where the responder thresholds are a direct result of the analyses described in the PAP. The process of deriving response definition values is described in brief in section 2.4.3.2. In section 2.4.2 the imputation approach for WOMAC (item) scores was clarified. In section 2.4.3 it was added that risk differences will be reported for binary endpoints. | Compliance with protocol and finalisation of the psychometric analysis report (PAP). |
| 5.0<br>(17 May 2023) | In the estimand description, the relevance of washout compliance intercurrent event was clarified for | Correspondence with the Food and Drug |
| | secondary endpoints. | Administration, US, has prompted further clarifications on |

SAP NN9536-4578 SAP | 5 of 28

Statistical Analysis Plan Trial ID: NN9536-4578

EudraCT No: 2017-003436-36


Date: Version: Status: Page:

13 November 2023 | Novo Nordisk

Final 6 of 28

The endpoint "Change in SF-36 general health score" has been moved from supportive secondary to exploratory in alignment with protocol.

Supportive secondary endpoint of "Change in pain medication" was changed to "Use of pain medication" to reflect descriptive character of the endpoint.

The calculation of WOMAC scores, including handling of partially missing assessments, has been clarified in details in section 2.4.1. In this section it was also clarified that SF-36 scores are norm based scores obtained from dedicated software.

In section 2.4.2 it has been clarified that the primary endpoint related to WOMAC is derived based on transformed and normalized WOMAC score as described in 2.4.1.

Prompted by FDA feedback, the decision on imputing data on the item level was retracted and it was clarified that missing WOMAC assessments will be imputed on the score level.

In section 2.4.2 additional sensitivity analysis was added for the primary endpoint of change in WOMAC pain score to address potential date/visit mismatch for 7 subjects.

Tables Table 2-4, Table 2-5, Table 2-7, Table 2-8 were added to give an overview of all planned analysis on all endpoints.

In section 2.4.3 it has been clarified that MMRM on endpoints related to WOMAC and SF-36 analysis addressing additional estimand will not use assessments not collected in compliance with the washout period for pain medication. In section 2.4.3.1 the description of analyses were updated to include the confirmatory secondary endpoint of change in SF-36 physical functioning.

In section 2.4.3.2 it was clarified that pain intensity (NRS) for each subject will be calculated as the mean of the available daily pain scores reported from 4 up to 7 days prior to the visit. The exclusion of data reported in washout period for pain intensity was done to facilitate interpretation of the results without imposed limitations on pain medication use. Additionally, it was noted that all endpoints derived from pain

WOMAC scores calculation (including handling of partially missing assessment).

SAP NN9536-4578 SAP of 28 Statistical Analysis Plan
Trial ID: NN9536-4578
Date: 13 November 2023 | Novo Nordisk
Version: 6.0

 Trial ID: NN9536-4578
 Version: Status: Final 

| | medication diary (use of pain medication and endpoints related to use of allowed rescue analgesics during washout period) will be analysed descriptively and descriptive statistics to be used were listed. Also, detailed definitions for deriving endpoints related to rescue analgesics from pain medication diary were specified. | |
|---|---|---|
| | The final thresholds are established based on FAS and prior to unblinding as per FDA request. This has been reflected in section 2.4.3.2 and the description of preliminary thresholds evaluation has been removed as no longer relevant. | |
| | A table <u>Table 2-6</u> summarising thresholds for meaningful within-patient change used in the PROs responder definitions was added in section 2.4.3.2. | |
| 6.0<br>(13 Nov 2023) | In section 2.4.2 the reduction procedure for imputation model was optimized and the description of further step in the procedure was added. | Corrections to imputation model reduction and imputation approach |
| | In section 2.4.3.1 the imputation approach for endpoints related to pain intensity (NRS) was changed to J2R-MI. | for endpoints related to pain intensity (NRS) were prompted by issues related to fitting the imputation model due to low availability of retrieved data for these endpoints. |

SAP NN9536-4578 SAP | 7 of 28

Statistical Analysis Plan
Trial ID: NN9536-4578


Date: 13 November 2023 Version: 6.0 Status: Final 

#### 1 Introduction

#### 1.1 Trial information

#### 1.1.1 Objective(s)

#### 1.1.1.1 Primary objective

To confirm superiority of semaglutide s.c. 2.4 mg once-weekly versus semaglutide placebo as an adjunct to a reduced-calorie diet and increased physical activity in subjects with obesity and knee OA in change from baseline to week 68 in body weight and knee OA-related pain.

#### 1.1.1.2 Secondary objectives

To confirm superiority of semaglutide s.c. 2.4 mg once-weekly versus semaglutide placebo as an adjunct to a reduced-calorie diet and increased physical activity in subjects with obesity and knee OA in achieving body weight response criteria after 68 weeks from baseline as well as change from baseline to week 68 in knee OA-related and general physical function.

To compare the efficacy of semaglutide s.c. 2.4 mg once-weekly versus semaglutide placebo as an adjunct to a reduced-calorie diet and increased physical activity in subjects with obesity and knee OA in change from baseline to week 68 in waist circumference, knee OA-related stiffness, overall knee OA-related physical limitations and general health-related quality of life.

#### 1.1.1.3 Exploratory objectives

To compare the efficacy of semaglutide s.c. 2.4 mg once-weekly versus semaglutide placebo as adjunct to a reduced-calorie diet and increased physical activity in subjects with obesity and knee OA in change from baseline to week 68 in use of analgesics and on walking distance.

#### 1.1.2 Estimands

#### 1.1.2.1 Primary estimand

The primary clinical question of interest is: what is the average treatment effect of semaglutide s.c. 2.4 mg once-weekly relative to semaglutide placebo as an adjunct to a reduced-calorie diet and increased physical activity, in patients with obesity and knee OA, measured by change from baseline to week 68 in body weight and knee OA-related pain, regardless of adherence to randomised treatment, regardless of initiating other anti-obesity therapies (weight management drugs or bariatric surgery) or other knee OA interventions (joint replacement or steroid injection or opioid medication) and regardless of compliance with washout period for pain medication (the latter only relevant in this context for knee OA-related pain) ("treatment policy" strategy).

The estimand is described by the following attributes (according to ICH E9(R1)):

- Treatment condition: The randomised treatment regardless of adherence or initiation of other anti-obesity therapies (as defined above) or other knee OA interventions (as defined above)
- Population: Patients with obesity and knee OA

Statistical Analysis Plan
Trial ID: NN9536-4578


Date: 13 November 2023 Version: 6.0
Status: Final


- Endpoints: The two primary endpoints relative change in body weight and change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score both from baseline to week 68
- Remaining intercurrent events: The intercurrent events "treatment discontinuation for any reason", "initiation of other anti-obesity therapies" and "initiation of other knee OA interventions" are addressed by the treatment condition attribute. The remaining intercurrent event is "compliance with washout period for pain medication" (in general only applicable to WOMAC endpoints), which is handled by the treatment policy strategy
- Population-level summary: Difference in mean changes between treatment conditions

A similar estimand applies to secondary endpoints (confirmatory, supportive) and exploratory endpoints related to body weight, waist circumference, WOMAC, SF-36 and pain intensity (NRS), which is called secondary estimand. The population-level summary for body weight response and WOMAC pain response endpoints is the ratio of odds between treatment conditions.

Rationale for estimand: The primary (and secondary) estimand was requested by different regulatory authorities and it aims at reflecting how patients with obesity are treated in clinical practice

#### 1.1.2.2 Additional estimand

An additional clinical question of interest is: what is the average treatment effect of semaglutide s.c. 2.4 mg once-weekly relative to semaglutide placebo as an adjunct to a reduced-calorie diet and increased physical activity, in patients with obesity and knee OA, measured by change from baseline to week 68 in body weight and knee OA-related pain, had they remained on their randomised treatment for the entire planned duration of the trial, not initiated other anti-obesity therapies (weight management drugs or bariatric surgery) or other knee OA interventions (joint replacement or steroid injection or opioid medication) and had they additionally complied with the washout period for pain medication (the latter only relevant in this context for knee OA-related pain) ("hypothetical" strategy).

The estimand is described by the following attributes (according to ICH E9(R1)):

- Treatment condition: The randomised treatment if patients had adhered for the entire duration of the trial, not initiated other anti-obesity therapies (as defined above) or other knee OA interventions (as defined above)
- Population: Patients with obesity and knee OA
- Endpoints: The two primary endpoints relative change in body weight and change in WOMAC pain score both from baseline to week 68
- Remaining intercurrent events: The intercurrent events "treatment discontinuation for any reason", "initiation of other anti-obesity therapies" and "initiation of other knee OA interventions" are addressed by the treatment condition attribute. The remaining intercurrent event is "compliance with washout period for pain medication" (in general only applicable to WOMAC endpoints), which is handled by the hypothetical strategy.
- Population-level summary: Difference in mean changes between treatment conditions

Statistical Analysis Plan
Trial ID: NN9536-4578
EudraCT No: 2017-003436-36

Status: Final 

A similar additional estimand applies to secondary endpoints (confirmatory and supportive) and exploratory endpoints related to body weight, waist circumference, WOMAC, SF-36 and pain intensity (NRS). The remaining intercurrent event of "compliance with washout period for pain medication" is considered relevant for all WOMAC and SF-36 related endpoints. The population-level summary for body weight response and WOMAC pain response endpoints is the ratio of odds between treatment conditions.

Rationale for estimand: The additional estimand was requested by few regulatory authorities and aims at reflecting the treatment effect in the absence of intercurrent events.

### 1.1.3 Endpoints

#### 1.1.3.1 Primary endpoints

| Endpoint title | Time frame | Unit |
|---|---|---|
| Change in body weight | From baseline (week 0) to end of treatment (week 68) | % |
| Change in WOMAC pain score | From baseline (week 0) to end of treatment (week 68) | Score points |

WOMAC; Western Ontario and McMaster Universities Osteoarthritis Index

#### 1.1.3.2 Confirmatory secondary endpoints

| Endpoint title | Time frame | Unit |
|---|---|---|
| Achieving body weight reduction | From baseline (week 0) to end of | Count of subject |
| ≥5% (yes/no) | treatment (week 68) | |
| Achieving body weight reduction ≥10% (yes/no) | From baseline (week 0) to end of treatment (week 68) | Count of subject |
| Change in WOMAC physical function score | From baseline (week 0) to end of treatment (week 68) | Score points |
| Change in SF-36 physical | From baseline (week 0) to end of | Score points |
| functioning score | treatment (week 68) | |

WOMAC; Western Ontario and McMaster Universities Osteoarthritis Index, SF-36; Short Form (36) Health Survey

## 1.1.3.3 Supportive secondary endpoints

| Endpoint title | Time frame | Unit |
|---|---|---|
| Change in waist circumference | From baseline (week 0) to end of treatment (week 68) | cm |
| Change in WOMAC stiffness score | From baseline (week 0) to end of treatment (week 68) | Score points |
| Change in WOMAC total score | From baseline (week 0) to end of treatment (week 68) | Score points |
| Change in SF-36 bodily pain score | From baseline (week 0) to end of treatment (week 68) | Score points |
| Change in SF-36 physical component summary | From baseline (week 0) to end of treatment (week 68) | Score points |
| Change in SF-36 mental component summary | From baseline (week 0) to end of treatment (week 68) | Score points |
| Use of allowed rescue analgesics during wash out | From baseline (week 0) to end of treatment (week 68) | Count of subjects |

SAP NN9536-4578 SAP | 10 of 28

| Statistical Analysis Plan | Date: | 13 November 2023 | Novo Nordisk |
|---|---|---|---|
| EudraCT No: 2017-003436-36 | Page: | 11 of 28 | |

| Amount of allowed rescue analgesics | From baseline (week 0) to end of | Dose |
|---|---|---|
| used during wash out | treatment (week 68) | |
| Use of pain medication | From baseline (week 0) to end of | Dose |
| | treatment (week 68) | |
| Change in pain intensity (NRS) | From baseline (week 0) to end of | Score points |
| | treatment (week 68) | |

WOMAC; Western Ontario and McMaster Universities Osteoarthritis Index, SF-36; Short Form (36) Health Survey

In addition to the protocol specified endpoints, the following supportive secondary endpoints are defined:

| Endpoint title | Time frame | Unit |
|---|---|---|
| Achieving body weight reduction | From baseline (week 0) to end of | Count of subject |
| ≥15% (yes/no) | treatment (week 68) | |
| Achieving body weight reduction ≥20% (yes/no) | From baseline (week 0) to end of treatment (week 68) | Count of subject |
| Achieving WOMAC pain reduction ≥30% (yes/no) | From baseline (week 0) to end of treatment (week 68) | Count of subject |
| Achieving WOMAC pain reduction ≥50% (yes/no) | From baseline (week 0) to end of treatment (week 68) | Count of subject |
| Achieving threshold(s) for clinically meaningful within-subject change in WOMAC pain score | From baseline (week 0) to end of treatment (week 68) | Count of subjects |
| Achieving threshold(s) for clinically meaningful within-subject change in WOMAC physical function score | From baseline (week 0) to end of treatment (week 68) | Count of subjects |
| Achieving threshold(s) for clinically meaningful within-subject change in SF-36 physical functioning score | From baseline (week 0) to end of treatment (week 68) | Count of subjects |
| Achieving pain intensity (NRS) reduction $\geq$ 30% (yes/no) | From baseline (week 0) to end of treatment (week 68) | Count of subject |
| Achieving pain intensity (NRS) reduction ≥50% (yes/no) | From baseline (week 0) to end of treatment (week 68) | Count of subject |

## 1.1.3.4 Exploratory endpoint(s)

| Endpoint title | Time frame | Unit |
|---|---|---|
| Change in 6 minutes walking | From baseline (week 0) to end of | Meters |
| distance | treatment (week 68) | |
| Change in SF-36 role-physical score | From baseline (week 0) to end of | Score points |
| | treatment (week 68) | |
| Change in SF-36 general health score | From baseline (week 0) to end of | Score points |
| | treatment (week 68) | |
| Change in SF-36 vitality score | From baseline (week 0) to end of | Score points |
| | treatment (week 68) | |
| Change in SF-36 social functioning | From baseline (week 0) to end of | Score points |
| score | treatment (week 68) | |
| Change in SF-36 role-emotional | From baseline (week 0) to end of | Score points |
| score | treatment (week 68) | |
| Change in SF-36 mental health score | From baseline (week 0) to end of | Score points |
| | treatment (week 68) | |

SAP NN9536-4578 SAP | 11 of 28

Statistical Analysis Plan
Trial ID: NN9536-4578
EudraCT No: 2017-003436-36

Date: 13 November 2023 | Novo Nordisk
Version: 6.0
Status: Final


#### 1.1.4 Type of trial

This is a 68-week, randomised, two-arm, double-blinded, multi-centre clinical trial comparing semaglutide s.c. 2.4 mg once-weekly with semaglutide placebo in subjects with moderate OA of one or both knees, pain due to knee OA, and obesity (BMI  $\geq$ 30.0 kg/m<sup>2</sup>).

### 1.2 Scope of the statistical analysis plan

This statistical analysis plan (SAP) is based on the updated protocol for trial NN9536-4578 "Effect of subcutaneous semaglutide 2.4 mg once-weekly compared to placebo in subjects with obesity and knee osteoarthritis", version 3.0 (21 April 2021) and includes more detailed procedures for executing the statistical analyses.

SAP NN9536-4578 SAP 12 of 28

13 November 2023 | Novo Nordisk Statistical Analysis Plan Date: Trial ID: NN9536-4578 Version: 6.0 CONFIDENTIA Final Status: EudraCT No: 2017-003436-36

Page:

13 of 28

#### 2 Statistical considerations

#### 2.1 Statistical hypotheses

The tests of superiority of semaglutide s.c. 2.4 mg once-weekly to semaglutide placebo for the two primary and all confirmatory secondary endpoints are performed using a fixed-sequence statistical strategy and a weighted Holm-Bonferroni procedure (with weights one). For a detailed specification of statistical hypotheses for the two primary endpoints see section 2.4.2.

This strategy tests the endpoints using a predefined hierarchical order; first the two primary endpoints: body weight change (%) and change in WOMAC pain score are tested at the significance level of 5% where the alpha is split between the two endpoints using 1% for body weight change (%) and 4% for change in WOMAC pain score.

If superiority is not confirmed for both endpoints, then the testing will stop. If the test of superiority for one of the two primary endpoints is significant, then the alpha can be recycled for the other primary endpoint, which will be tested at the 5% significance level. If both hypotheses are rejected and superiority is confirmed, then the confirmatory secondary endpoints (starting with  $\geq 5\%$  body weight reduction) will be tested at the 5% level. Testing for superiority of confirmatory secondary endpoints can proceed only after a statistically significant result (p-value < 5%) on the previous endpoint.

#### 2.2 Sample size determination

The trial is designed with an effective power of 90% and 67% to detect differences on the two primary endpoints and confirmatory secondary endpoints, respectively. The effective power was calculated under the assumption of independence of endpoints by multiplying the respective marginal powers successively which is a conservative approach. The power calculations for continuous endpoints are based on a t-test on the mean difference assuming equal variances, whereas those for the categorical endpoints are based on the Pearson chi-square test for two independent proportions.

Assumptions for these calculations are presented in Table 2-1 and are based on findings from NN9536-4153 and NN9536 phase 3a program (STEP) as well as on relevant publications on body weight loss and knee OA outcome (using WOMAC). Two studies, Bliddal et al. and Christensen et al., found that weight loss treatment (average weight loss 7.5% and 6.8% respectively) could lead to improvements in knee OA symptoms like pain and physical function (pain score: -8.4 (-10.4 vs -2.0) with baseline score 38.4 (SD=21.1) and -5.4 (-11.4 vs -6.0) with baseline score 36.7 (SD=21.3) respectively; function score: -3.7 (-10.2 vs -6.5) with baseline score 39.2 (SD=21.4) and -9.9 (-14.9 vs -5.0) with baseline value 37.4 (SD=21.8) respectively) in obese subjects (average BMI at baseline 35.6 and 35.9 respectively)<sup>4.5</sup>. Aforementioned score improvements were found in treatment completers. Item responses were collected using the visual analogue scale (VAS) format of the questionnaire. Bliddal et al. reported normalised sum of scores (range 0-100) and Christensen et al. reported sum of scores, which were transformed to a 0-100 range for comparison purposes. Consequently, a treatment difference for the pain score was assumed to be -9 (-11 vs -2) with SD=20; for the function score it was assumed to be -9 (-15 vs -6) with SD=19 if treated with semaglutide s.c. 2.4 mg once-weekly vs semaglutide placebo for 68 weeks. Clement et al. identified a minimum clinically important difference of 11 for pain and 9 for function and a minimum

13 SAP NN9536-4578 SAP of 28 Statistical Analysis Plan
Trial ID: NN9536-4578
EudraCT No: 2017-003436-36

Status: Final 

important change of 21 for pain and 16 for function for improvement in WOMAC after total knee arthroplasty. Although, it is planned to use the numerical rating scale (NRS) format of the questionnaire in this trial, it is known that VAS and NRS are highly correlated (r>0.93) and that VAS derived assumptions for sample size calculation are adequate and can be translated to a setting where NRS is used. It is planned that the WOMAC scores (derived from NRS responses) will be transformed to a 0-100 range based on which the corresponding endpoints will be calculated.

In relation to expected treatment effects it was assumed that 20% of subjects discontinue permanently and 60% of these are retrieved at week 68. All subjects in the placebo arm are assumed to have same effect as subjects who complete the trial on placebo. Retrieved subjects in the semaglutide s.c. 2.4 mg once-weekly arm are assumed to have an effect corresponding to half the treatment difference (compared to placebo) of subjects who complete the trial on semaglutide s.c. 2.4 mg once-weekly. Non-retrieved subjects in the semaglutide s.c. 2.4 mg once-weekly arm are assumed to have an effect corresponding to placebo.

Under these assumptions and a 2:1 randomisation ratio, the desired power of at least 90% for change in WOMAC pain score is obtained with 375 subjects randomised to either receive semaglutide s.c. 2.4 mg once-weekly (250) or placebo (125).

Table 2-1 Assumptions, marginal power and effective power for each endpoint in the hierarchical testing procedure given an anticipated number of 375 randomised subjects

| Order | Endpoint | Assumed mo | ean (±SD) or<br>or completers | Expected<br>mean (±SD)<br>or<br>proportion | Expected difference or | Marginal<br>power | Two-sided<br>significance | |
|---|---|---|---|---|---|---|---|---|
| | | Semaglutide<br>s.c. 2.4 mg<br>once-weekly | Semaglutide<br>placebo | Semaglutide<br>s.c. 2.4 mg<br>once-weekly | proportion<br>ratio | (%) | level (%) * | (%) |
| 1 | % body<br>weight<br>change # | 14.0 (±10) | 3.0 (±10) | 12.5 (±11) | 9.5%-<br>points | >99 | 1 | 99 |
| 1 | WOMAC<br>pain change<br># | 11.0 (±20) | 2.0 (±20) | 9.7 (±21) | 7.7 score-<br>points | 90 | 4 | 90 |
| 2 | 5% responders | 82% | 42% | 76% | 1.8 | >99 | 5 | 90 |
| 3 | 10%<br>responders | 66% | 24% | 60% | 2.5 | >99 | 5 | 90 |
| 4 | WOMAC function change # | 15.0 (±19) | 6.0 (±19) | 13.7 (±20) | 7.7 score-<br>points | 94 | 5 | 84 |
| 5 | SF-36<br>physical<br>functioning<br>change | 6.0 (±10) | 2.0 (±10) | 5.4 (±11) | 3.4 score-<br>points | 80 | 5 | 67 |

SD: Standard deviation; WOMAC: Western Ontario McMasters Osteoarthritis Index ; SF-36: Short Form (36) Health Survey.

<sup>\*</sup>Significance level for confirmatory secondary endpoints reflects local alpha if all superiority hypotheses for endpoints higher in the statistical hierarchy were rejected

Statistical Analysis Plan
Trial ID: NN9536-4578
EudraCT No: 2017-003436-36

Status: Final 

# Shown as a positive number

As currently there are no Novo Nordisk trials utilising WOMAC, see <u>Table 2-2</u> for alternative power calculations to the main scenario assuming varying sample size, mean difference or standard deviation.

Table 2-2 Marginal power for WOMAC pain change (shown as a positive number) for alternative sample size, mean difference or standard deviation

| Sample size | Expected mean<br>for semaglutide<br>placebo | Expected mean<br>for semaglutide<br>s.c. 2.4 mg once-<br>weekly | Expected difference | Common SD | Marginal<br>power (%) |
|---|---|---|---|---|---|
| Main scenario | | Weekiy | 1 | | |
| 375 | 2 | 9.7 | 7.7 | 21 | 0.900 |
| Varying sample | size | · I | | l . | l . |
| 285 | 2 | 9.7 | 7.7 | 21 | 0.803 |
| 303 | 2 | 9.7 | 7.7 | 21 | 0.828 |
| 324 | 2 | 9.7 | 7.7 | 21 | 0.853 |
| 348 | 2 | 9.7 | 7.7 | 21 | 0.877 |
| 375 | 2 | 9.7 | 7.7 | 21 | 0.900 |
| 411 | 2 | 9.7 | 7.7 | 21 | 0.925 |
| 462 | 2 | 9.7 | 7.7 | 21 | 0.951 |
| 543 | 2 | 9.7 | 7.7 | 21 | 0.975 |
| 888 | 2 | 9.7 | 7.7 | 21 | >.999 |
| Varying mean d | ifference | • | 1 | 1 | |
| 375 | 2 | 5 | 3 | 21 | 0.226 |
| 375 | 2 | 6 | 4 | 21 | 0.375 |
| 375 | 2 | 7 | 5 | 21 | 0.545 |
| 375 | 2 | 8 | 6 | 21 | 0.708 |
| 375 | 2 | 9 | 7 | 21 | 0.837 |
| 375 | 2 | 10 | 8 | 21 | 0.921 |
| 375 | 2 | 11 | 9 | 21 | 0.968 |
| 375 | 2 | 12 | 10 | 21 | 0.989 |
| 375 | 2 | 13 | 11 | 21 | 0.997 |
| 375 | 2 | 14 | 12 | 21 | >.999 |
| 375 | 2 | 15 | 13 | 21 | >.999 |
| Varying standar | rd deviation | | | | |
| 375 | 2 | 9.7 | 7.7 | 10 | >.999 |
| 375 | 2 | 9.7 | 7.7 | 11 | >.999 |
| 375 | 2 | 9.7 | 7.7 | 12 | >.999 |
| 375 | 2 | 9.7 | 7.7 | 13 | >.999 |
| 375 | 2 | 9.7 | 7.7 | 14 | 0.998 |
| 375 | 2 | 9.7 | 7.7 | 15 | 0.996 |
| 375 | 2 | 9.7 | 7.7 | 16 | 0.990 |
| 375 | 2 | 9.7 | 7.7 | 17 | 0.981 |
| 375 | 2 | 9.7 | 7.7 | 18 | 0.967 |
| 375 | 2 | 9.7 | 7.7 | 19 | 0.949 |
| 375 | 2 | 9.7 | 7.7 | 20 | 0.927 |
| 375 | 2 | 9.7 | 7.7 | 21 | 0.900 |

SAP NN9536-4578 SAP 15 of 28

| Statistical Analyst<br>Trial ID: NN953<br>EudraCT No: 20 | 6-4578 | CONF | I <del>DENTIAL</del> | Date:<br>Version:<br>Status:<br>Page: | 13 November 2023 <b>Novo Nordisk</b> 6.0 Final 16 of 28 |
|---|---|---|---|---|---|
| 375 | 2 | 9.7 | 7.7 | 22 | 0.871 |
| 375 | 2 | 9.7 | 7.7 | 23 | 0.840 |
| 375 | 2 | 9.7 | 7.7 | 24 | 0.807 |
| 375 | 2 | 9.7 | 7.7 | 25 | 0.773 |
| 375 | 2 | 9.7 | 7.7 | 26 | 0.740 |
| 375 | 2 | 9.7 | 7.7 | 27 | 0.706 |
| 375 | 2 | 9.7 | 7.7 | 28 | 0.673 |
| 375 | 2 | 9.7 | 7.7 | 29 | 0.642 |
| 375 | 2 | 9.7 | 7.7 | 30 | 0.611 |

SD: Standard deviation.

All above outlined sample size and power considerations are for the primary estimand for primary endpoints or the secondary estimand for confirmatory secondary endpoints (treatment policy strategy). It is assumed that up to 20% of subjects discontinue permanently and 60% of these are retrieved at week 68, which amounts to 8% expected missing data at week 68. Based on NN9536 STEP 1 trial 8.8% missing in-trial data was observed after 68 weeks for the primary estimand. Any superiority conclusions will be based on the primary or secondary estimand.

For the additional estimand (hypothetical strategy) however, data from retrieved subjects are not used. Hence, it is expected that up to 20% of data will be missing at week 68. Based on NN9536 STEP 1 trial 20.6% missing on-treatment data was observed after 68 weeks for the additional estimand. This included missing data not only due to treatment discontinuation, but also due to initiation of other anti-obesity therapies (<1%). For trial NN9536-4578 slightly higher missing ontreatment data is expected due to subjects initiating other knee OA interventions (<3%) and not complying with the washout period (<10%). In NN9536 STEP 1 trial it was seen that the treatment difference in mean changes for body weight was slightly higher and standard deviation was slightly lower for the additional estimand (using on-treatment data) than for the primary estimand (using intrial data).

#### 2.3 Definition of analysis sets

Two analysis sets are defined:

The *full analysis set* (*FAS*) includes all randomised subjects according to the intention-to-treat principle. The subjects in the *FAS* contribute to the evaluation as randomised.

The *safety analysis set (SAS)* includes all randomised subjects exposed to at least one dose of randomised treatment. The subjects in the *SAS* contribute to the evaluation as treated.

Any observation excluded from the analysis database will be documented before database lock with the reason for exclusion provided. Efficacy endpoints will be analysed using the FAS; safety endpoints will be analysed using the SAS.

Two observation periods are defined for each subject:

In-trial: The *in-trial period* is defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site.

SAP NN9536-4578 SAP | 16 of 28

| Statistical Analysis Plan | Date: | 13 November 2023 | Novo Nordisk |
|---|---|---|---|
| EudraCT No: 2017-003436-36 | Page: | 17 of 28 | |

On-treatment (with trial product): A time-point is considered as "on-treatment" if any dose of trial product has been administered within the prior 2 weeks (14 days). The *on-treatment period* is defined as all times which are considered on-treatment.

In general, the *on-treatment period* will therefore be from the date of first trial product administration to date of last trial product administration excluding potential off-treatment time intervals triggered by at least two consecutive missed doses.

For the evaluation of AEs, the lag time for each on-treatment time interval is 7 weeks (49 days).

The in-trial and on-treatment periods define the patient years of observation (PYO) and patient years of exposure (PYE), respectively, as the total time duration in the periods.

#### 2.4 Statistical analyses

#### 2.4.1 General considerations

The last available and eligible observation at or before randomisation is used as the baseline value. If no assessments are available, the mean value at randomisation across all subjects is used as the baseline value.

#### **WOMAC** scores considerations

The WOMAC raw pain score is derived as the sum of the 5 item scores in the pain domain. The WOMAC raw physical function score is derived as the sum of the 17 item scores in the physical function domain. The WOMAC raw stiffness score is derived as the sum of the 2 item scores in the stiffness domain. The WOMAC raw total score is derived as the sum of all 24 item scores.

All WOMAC raw scores (domain scores and total score) will be normalised and expressed on a 0-100 scale. This is done by dividing raw score by the highest possible value of the raw score for the domain (see <u>Table 2-3</u>) and multiplying by 100.

#### Handling partially missing responses

In the event of missing items the response for the domain can still be considered valid. The minimal numbers of available items required per domain for the score to be calculated from the data are presented in the <u>Table 2-3</u>. If the number of available items criterium for the domain score validity is not met, the raw score cannot be calculated and is considered missing. Otherwise the raw score is calculated as an average of the available items and multiplied by number of all items in the domain. The total score is calculated from the data only if all 3 domain scores are valid.

SAP NN9536-4578 SAP | 17 of 28

13 November 2023 Novo Nordisk Statistical Analysis Plan Date: Trial ID: NN9536-4578 Version: CONFIDENTIAL

Final Status: EudraCT No: 2017-003436-36 18 of 28 Page:

6.0



#### SF-36 scores considerations

The SF-36 composite scores used to calculate corresponding endpoints are norm based scores (NBS) and will be obtained from PRO-CoRE software by QualityMetric.

#### 2.4.2 Primary endpoint(s)

The primary endpoints are change in body weight (%) and change in WOMAC pain score from baseline (week 0) to end of treatment (week 68) as listed in section 3 of the protocol. Regarding WOMAC, then the version used is the WOMAC 3.1 NRS version, an 11-point numeric rating scale with responses ranging from no symptom/difficulty (0) to extreme symptom/difficulty (10). The version has a 24-hour recall period.

Change from baseline to week 68 in body weight (%) is defined as

% body weight change = 
$$\frac{\text{(body weight at week 68 - body weight at baseline)}}{\text{body weight at baseline}} \times 100.$$

Change from baseline to week 68 in WOMAC pain score is defined as

WOMAC pain score change = WOMAC pain score at week 68 – WOMAC pain score at baseline,

where the WOMAC pain score is the transformed raw score, that is, normalised and represented on a scale of 0-100, as described in 2.4.1.

All tests are tests of superiority of semaglutide s.c. 2.4 mg once-weekly to semaglutide placebo.

18 of 28 SAP NN9536-4578 SAP

| Statistical Analysis Plan | Date: | 13 November 2023 | Novo Nordisk |
|---|---|---|---|
| EudraCT No: 2017-003436-36 | Page: | 19 of 28 | |

Let  $\mu_{semaglutide}$  and  $\mu_{semaglutide}$  denote the true mean of % body weight change or WOMAC pain score change for semaglutide s.c. 2.4 mg once-weekly and semaglutide placebo, respectively. The null and alternative hypotheses tested are

```
H_0: \mu_{semaglutide} \ge \mu_{semaglutide \ placebo} \ vs

H_A: \mu_{semaglutide} < \mu_{semaglutide \ placebo}.
```

The null hypotheses will be rejected and superiority claimed, if the obtained p-value is below the significance level on which the testing is performed and the direction of the estimated effect favours semaglutide.

#### Analyses addressing the primary estimand

The following statistical analyses and imputation methods are designed to address the primary estimand.

The analysis model for change in body weight (%) and change in WOMAC pain score will be a linear regression (ANCOVA) with randomised treatment as factor and either baseline body weight (kg) or baseline WOMAC pain score as covariate assuming equal variances. The estimated treatment difference between semaglutide s.c. 2.4 mg once-weekly and semaglutide placebo will be reported together with the associated two-sided 95% confidence interval (CI) and corresponding p-value.

Body weight measurements and WOMAC pain scores that are missing at week 68 will be imputed based on available data at week 68 and the endpoint will be derived from the imputed values, i.e. % body weight change and WOMAC pain score change.

Multiple imputation approach using retrieved subjects (RD-MI): The primary imputation approach for the primary estimand is a multiple imputation similar to the one described by McEvoy1. For subjects in the semaglutide s.c. 2.4 mg once-weekly and the semaglutide placebo arms, missing measurements at week 68 for non-retrieved subjects are imputed using all available week 68 assessments from retrieved subjects in each randomised treatment arm. This will be done according to the timing of last available observation during the on-treatment period (LAO-OT) as well as by taking sex, baseline BMI and baseline body weight / WOMAC pain score into account. Missing measurements at week 68 for subjects on randomised treatment (at week 68) are imputed by sampling from available measurements at week 68 from subjects on randomised treatment in the relevant randomised treatment arms. The multiple imputation approach is done in three steps:

• Imputation: Defines an imputation model using retrieved subjects from FAS and done within groups defined by randomised treatment and end of treatment status (on-drug/off-drug). The model will be a linear regression of body weight (kg) / WOMAC pain score at week 68 with sex (male/female), baseline BMI (kg/m²) (in categories -<35, 35-<40, ≥40) and baseline body weight (kg) / WOMAC pain score, timing of last available observation during the on-treatment period (LAO-OT) and LAO-OT of body weight (kg) / WOMAC pain score as covariates. If no LAO-OT exists post-baseline then the LAO-OT will be the baseline body weight / WOMAC pain score and the timing will be 0. No interactions will be included. If the imputation model cannot be fit due to small group size, the model will be reduced until the model can be fit. Reduction will be done in a fixed order by first collapsing the two highest baseline BMI groups

SAP NN9536-4578 SAP | 19 of 28

Statistical Analysis Plan
Trial ID: NN9536-4578
EudraCT No: 2017-003436-36

Status: Final 

into one (≥35), then removing baseline BMI group and finally removing sex. If the model still cannot be fit, the imputation will be done regardless of the randomised treatment arm. If no LAO-OT exists post-baseline then the LAO-OT will be the baseline body weight / WOMAC pain item score and the timing will be 0. The estimated posterior distribution for the parameters (regression coefficients and variances) in the imputation models are then used to impute missing week 68 body weight / WOMAC pain score values for each randomised treatment arm. This will be done 1,000 times and results in 1,000 complete data sets.

- **Analysis**: Analysis of each of the 1,000 complete data sets, using the analysis models (ANCOVA and logistic regression) results in 1,000 times 2 estimations.
- **Pooling**: Integrates the 1,000 times 2 estimation results into two final results using Rubin's formula.

Based on NN9536-4153 phase 2 results 1,000 copies should be sufficient to establish stable results. If 1,000 copies are insufficient, 10,000 copies will be used. The multiple imputations will be generated using Novo Nordisk trial number 95364578 as seed number. In addition to the seed number, it is specified that the dataset is sorted by subject ID.

#### Sensitivity analyses

Jump to reference multiple imputation approach (J2R-MI): Missing values of body weight / WOMAC pain score at week 68 for both the semaglutide 2.4 mg and semaglutide placebo group are imputed by sampling among all available assessments at week 68 in the semaglutide placebo group. This approach makes the assumption that subjects instantly after discontinuation lose any effect of randomised treatment beyond what can be expected from semaglutide placebo treatment as adjunct to reduced-calorie diet and increased physical activity2. The multiple imputation approach is done as above with the first step replaced by

• Imputation: Defines an imputation model using semaglutide placebo subjects from FAS with a week 68 measurement. The model will be a linear regression of body weight (kg) / WOMAC pain score at week 68 with sex (male/female), BMI (kg/m²) (in categories -<35, 35-<40, ≥40 as factors and baseline body weight (kg) / WOMAC pain score as covariate. No interactions will be included. If the imputation model cannot be fit due to inadequate numbers of retrieved subjects in 1 or more groups, then the imputation model will be reduced until the model can be fit. Reduction will be done in a fixed order by first collapsing the two highest baseline BMI-groups into one (≥35), then removing baseline BMI-group and finally removing sex. The estimated posterior distribution for the parameters (regression coefficients and variances) in the imputation models are then used to impute missing week 68 body weight / WOMAC pain score values for each randomised treatment arm. This will be done 1,000 times and results in 1,000 complete data sets.

Tipping-point multiple imputation analysis (TP-MI): First, missing data are imputed according to the primary multiple imputation approach. Then, a penalty is added to the imputed values at week 68. The approach is to explore a range of penalties for both treatment groups, and the impact these would have on the study conclusions. The 2-dimensional space of penalties covering the range from -30% to 30% (for body weight change) / -50 to 50 (for WOMAC pain score) will be explored for both treatment groups. This sensitivity analysis evaluates the robustness of the superiority

SAP NN9536-4578 SAP 20 of 28

Statistical Analysis Plan
Trial ID: NN9536-4578
EudraCT No: 2017-003436-36

Status: Final 

conclusions to departures from the observed change in body weight / WOMAC pain score in both treatment groups.

ANCOVA for unequal variances: An alternative analysis model similar to the primary analysis model (ANCOVA), following the primary imputation approach (RD-MI), but assuming unequal variances instead of equal variances. The analysis model includes randomised treatment as factor and either baseline body weight (kg) or baseline WOMAC pain score as covariate. The estimated treatment difference between semaglutide s.c. 2.4 mg once-weekly and semaglutide placebo will be reported together with the associated two-sided 95% confidence interval (CI) and corresponding p-value.

ANCOVA addressing date/visit mismatch: This sensitivity analysis uses the same analysis model and imputation approach as the primary analysis, and aims to evaluate the robustness of the results for the primary endpoint of change in WOMAC pain score to potential data issues for 7 subjects (subject ids: 455005, 551016, 611003, 614003, 614011, 614012, 614013) for whom there is a mismatch between the WOMAC assessment date and assigned visit that impacts the primary endpoint derivation at week 68. The assessments in question will be reassigned to the visit matching the assessment date.

#### Analyses addressing the additional estimand

The additional estimand for change in body weight (%) and change in WOMAC pain score will be assessed using a mixed model for repeated measurements (MMRM) approach.

Week 68 assessments for retrieved subjects are not used in this analysis. The MMRM will use assessments only from subjects who are taking the randomised treatment until end of treatment or until first discontinuation of randomised treatment. For subjects who experience other intercurrent events before completion or first discontinuing of randomised treatment, the date of initiating other anti-obesity therapies (weight management drugs or bariatric surgery) or other knee OA interventions (joint replacement or steroid injections) will be used as latest date for using assessments in this MMRM. Additionally, for the MMRM analysing change in WOMAC pain score, assessments not collected in compliance with the washout period for pain medication will not be used. The MMRM will be fitted using the change (% body weight change or change in WOMAC pain score) and the same factor and covariate as for the primary analysis all nested within visit. An unstructured covariance matrix for measurements within the same subject will be employed, assuming that measurements for different subjects are independent.

SAP NN9536-4578 SAP 21 of 28

| Statistical Analysis Plan | Date: | 13 November 2023 | Novo Nordisk |
|---|---|---|---|

| CONFIDENTIAL | Status: | Final | Page: | 22 of 28 |

Table 2-4 Analysis and imputation methods to address the primary and additional estimands for primary endpoints

| Endpoint title | Unit | Endpoint | Strategy | Analysis set | Statistical model | Imputation approach | Sensitivity analysis |
|---|---|---|---|---|---|---|---|
| Change in body weight | % | Continuous | Treatment policy | FAS | ANCOVA | RD-MI | J2R-MI<br>TP-MI<br>Uneq.Var. |
| | | | Hypothetical | FAS | MMRM | - | - |
| Change in<br>WOMAC pain<br>score | Score points | Continuous | Treatment policy | FAS | ANCOVA | RD-MI | J2R-MI<br>TP-MI<br>Uneq.Var. |
| 50010 | | | Hypothetical | FAS | MMRM | - | - |

#### 2.4.3 Secondary endpoints

#### 2.4.3.1 Confirmatory secondary endpoints

Confirmatory secondary endpoints are listed in section <u>1.1.3.2</u>. All tests are tests of superiority of semaglutide s.c. 2.4 mg once-weekly to semaglutide placebo.

Table 2-5 Analysis and imputation methods to address the secondary and additional estimands for confirmatory secondary endpoints

| Endpoint title | Unit | Endpoint | Strategy | Analysis<br>set | Statistical model | Imputation approach | |
|---|---|---|---|---|---|---|---|
| Achieving body | Count of | D. | Treatment policy | FAS | LR | RD-MI | |
| weight reduction<br>≥5% (yes/no) | subject | Binary | Hypothetical | FAS | LR | MMRM | |
| Achieving body | Count of | D. | Treatment policy | FAS | LR | RD-MI | |
| weight reduction<br>≥10% (yes/no) | subject | Binary | Hypothetical | FAS | LR | MMRM | |
| Change in WOMAC | Score points | Score | G i | Treatment policy | FAS | ANCOVA | RD-MI |
| physical function score | | Continuous | Hypothetical | FAS | MMRM | - | |
| Change in SF-36 | Score | G .: | Treatment policy | FAS | ANCOVA | RD-MI | |
| physical functioning score points | Continuous | Hypothetical | FAS | MMRM | - | | |

#### Analyses addressing the secondary estimand

The confirmatory secondary endpoints addressing the secondary estimand will be analysed in a similar way as the primary endpoints addressing the primary estimand.

The statistical model for continuous confirmatory secondary endpoints will be the same linear regression as for the primary endpoints (ANCOVA) with treatment as a factor and the baseline value of the endpoint as covariate. The statistical model for confirmatory body weight responder endpoints is a logistic regression using randomised treatment as a factor and baseline body weight (kg) as covariate. The estimated odds ratio (OR) as well as risk differences between semaglutide s.c.

| Statistical Analysis Plan | Date: | 13 November 2023 | Novo Nordisk |
|---|---|---|---|
| EudraCT No: 2017-003436-36 | Page: | 23 of 28 | |

2.4 mg once-weekly and semaglutide placebo will be reported together with the associated two-sided 95% confidence interval and corresponding p-value.

The imputation approach is the same multiple imputation using retrieved subjects as described in section 2.4.2.

#### Analyses addressing the additional estimand

The confirmatory secondary endpoints change in WOMAC physical function score and change in SF-36 physical functioning score addressing the additional estimand will be analysed using the same MMRM as described for the primary endpoints addressing the additional estimand with randomised treatment as a factor and the baseline value of the endpoint as covariate. For these analyses assessments not collected in compliance with the washout period for pain medication will not be used.

The confirmatory body weight responder endpoints addressing the additional estimand will be analysed using the same MMRM described for the primary endpoint change in body weight (%) addressing the additional estimand except that body weight (kg) will be used as response variable in the model. For subjects with missing body weight at week 68, individual values for body weight will be predicted from the MMRM and used to classify each subject as 5% or 10% responder or not. This classification will then be analysed using a logistic regression model with randomised treatment as a factor and baseline body weight (kg) as covariate.

## 2.4.3.2 Supportive secondary endpoints

Supportive secondary endpoints are listed in section <u>1.1.3.3</u>. All tests are tests of superiority of semaglutide s.c. 2.4 mg once-weekly to semaglutide placebo.

## Analyses addressing the secondary estimand

The supportive secondary endpoints related to body weight, waist circumference, WOMAC and SF-36 addressing the secondary estimand will be analysed using the same imputation approach as used for the primary endpoints while supportive secondary endpoints related to pain intensity (NRS) will be analysed using the J2R-MI imputation approach as described for the sensitivity analysis of the primary endpoints. The statistical model for continuous endpoints will be the same linear regression as for the primary endpoints (ANCOVA) with treatment as a factor and the baseline value of the endpoint as covariate. The statistical model for responder endpoints is a logistic regression using treatment as a factor and baseline value of the endpoint as covariate. The estimated odds ratio (OR) as well as risk differences between semaglutide s.c. 2.4 mg once-weekly and semaglutide placebo will be reported together with the associated two-sided 95% confidence interval and corresponding p-value.

The baseline pain intensity (NRS) for each subject will be calculated as the mean of the available daily pain scores reported from 4 and up to 7 days prior to the randomisation visit. The means at each post-baseline visit until week 68 will be calculated in a similar way.

#### Analyses addressing the additional estimand

The supportive secondary endpoints related to body weight, waist circumference, WOMAC, SF-36, and pain intensity (NRS) addressing the additional estimand will be analysed using the same

SAP NN9536-4578 SAP | 23 of 28

Statistical Analysis Plan
Trial ID: NN9536-4578

Status: Final


MMRM as described for the primary endpoints addressing the additional estimand with randomised treatment as a factor and the baseline value of the endpoint as covariate. For the MMRM analysing endpoints related to WOMAC and SF-36, assessments not collected in compliance with the washout period for pain medication will not be used.

Responder endpoints (body weight, WOMAC pain or pain intensity (NRS)) addressing the additional estimand will be analysed using the same MMRM as described for the primary endpoint change in body weight (%) addressing the additional estimand except that the endpoint will be used as response variable in the model. For subjects with missing assessments at week 68, individual values will be predicted from the MMRM and used to classify each subject as a responder or not. This classification will then be analysed using a logistic regression model with randomised treatment as a factor and baseline value of the endpoint as covariate.

#### Other analyses

Use of pain medication and endpoints related to use of allowed rescue analgesics during washout period will be described using plots and descriptive statistics. Use of pain medication will be categorised into opioids, NSAIDs and acetaminophen. The summaries and plots will be done by these categories and will include overall time on medication, pain medication rates and prevalence plots. For opioids, time to event plot will be presented. The allowed rescue analgesics will be identified as acetaminophen reported in the pain medication diary 1, 2 or 3 days prior to WOMAC assessment and the individual amount of rescue analgesics at each visit will be calculated as a total dose reported taken on those days.

Responder analyses for WOMAC pain, WOMAC physical function and SF-36 physical functioning will be carried out with thresholds for clinically meaningful within-subject change derived prior to unblinding from NN9536-4578 data using anchor based methods (Patient Global Impression of Status and Patient Global Impression of Change items). The responder thresholds were derived by an external vendor based on the complete dataset prior to DBL. Responder analyses will be carried out on a range of responder thresholds including the final primary response definition values of clinically meaningful within-subject change for WOMAC pain, WOMAC physical function and SF-36 physical functioning based on one category improvement on the corresponding PGI-S items, plus the next lower/upper response value representing, respectively, no change and two category change on the PGI-S scale. The final thresholds are summarised in Table 2-6.

Table 2-6 Summary of the derived thresholds for meaningful within-subject change

| PGI-S group | WOMAC pain score | WOMAC physical | SF-36 physical |
|---|---|---|---|
| | | function score | functioning score |
| No change | -17.8 | -21.7 | 5.2 |
| 1-category improvement* | -37.3 | -41.2 | 11.4 |
| 2-category improvement | -53.0 | -49.8 | 16.4 |

<sup>\*)</sup> The derived threshold value for final primary response value of clinically meaningful within-subject change

Statistical Analysis Plan Date: 13 November 2023 November

 Trial ID: NN9536-4578
 Version: Status: Final 

Table 2-7 Analysis and imputation methods to address the secondary and additional estimands for supportive secondary endpoints

| Endpoint title | Unit | Endpoint | Strategy | Analysis set | Statistical model | Imputation approach |
|---|---|---|---|---|---|---|
| Change in waist | | Cti | Treatment policy | FAS | ANCOVA | RD-MI |
| circumference | cm | Continuous | Hypothetical | FAS | MMRM | - |
| Change in WOMAC | Score | Cantinuana | Treatment policy | FAS | ANCOVA | RD-MI |
| stiffness score | points | Continuous | Hypothetical | FAS | MMRM | - |
| Change in WOMAC | Score | Continuous | Treatment policy | FAS | ANCOVA | RD-MI |
| total score | points | Continuous | Hypothetical | FAS | MMRM | - |
| Change in SF-36 bodily | Score | Continuous | Treatment policy | FAS | ANCOVA | RD-MI |
| pain score | points | Continuous | Hypothetical | FAS | MMRM | - |
| Change in SF-36 | Score | Continuous | Treatment policy | FAS | ANCOVA | RD-MI |
| general health score | points | Continuous | Hypothetical | FAS | MMRM | - |
| Change in SF-36 | Score | | Treatment policy | FAS | ANCOVA | RD-MI |
| physical component<br>summary | points | Continuous | Hypothetical | FAS | MMRM | - |
| Change in SF-36 | Score | | Treatment policy | FAS | ANCOVA | RD-MI |
| mental component summary | points | Continuous | Hypothetical | FAS | MMRM | - |
| Use of allowed rescue<br>analgesics during wash<br>out | Count of subjects | Binary | - | FAS | Descriptive statistics | - |
| Amount of allowed rescue analgesics used during wash out | Dose | Continuous | - | FAS | Descriptive statistics | - |
| Use of pain medication | Number of days | Continuous | - | FAS | Descriptive statistics | - |
| Change in pain | Score | C · | Treatment policy | FAS | ANCOVA | J2R-MI |
| intensity (NRS) | points | Continuous | Hypothetical | FAS | MMRM | - |
| Achieving body weight | Count of | | Treatment policy | FAS | LR | RD-MI |
| reduction ≥15%<br>(yes/no) | subject | Binary | Hypothetical | FAS | LR | MMRM |
| Achieving body weight | Count of | | Treatment policy | FAS | LR | RD-MI |
| reduction ≥20%<br>(yes/no) | subject | Binary | Hypothetical | FAS | LR | MMRM |
| Achieving WOMAC | Count of | | Treatment policy | FAS | LR | RD-MI |
| pain reduction ≥30%<br>(yes/no) | subject | Binary | Hypothetical | FAS | LR | MMRM |

Statistical Analysis Plan
Trial ID: NN9536-4578
EudraCT No: 2017-003436-36

Status: Final 

| Endpoint title | Unit | Endpoint | Strategy | Analysis set | Statistical model | Imputation approach |
|---|---|---|---|---|---|---|
| Achieving WOMAC pain reduction ≥50% | Count of | Dinomy | Treatment policy | FAS | LR | RD-MI |
| yes/no) | subject | Binary | Hypothetical | FAS | LR | MMRM |
| Achieving threshold(s) for clinically meaningful | Count of | | Treatment policy | FAS | LR | RD-MI |
| within-subject change* in WOMAC pain score | subject | Binary | Hypothetical | FAS | LR | MMRM |
| Achieving threshold(s) | | | Treatment policy | FAS | LR | RD-MI |
| for clinically meaningful<br>within-subject change* in<br>WOMAC physical<br>function score | Count of subject | Binary | Hypothetical | FAS | LR | MMRM |
| Achieving threshold(s) for clinically meaningful | | | Treatment policy | FAS | LR | RD-MI |
| within-subject change* in SF-36 physical functioning score | Count of subject | Binary | Hypothetical | FAS | LR | MMRM |
| Achieving pain intensity | Count of | Dinomy | Treatment policy | FAS | LR | J2R-MI |
| (NRS) reduction ≥30%<br>(yes/no) | subject | Binary | Hypothetical | FAS | LR | MMRM |
| Achieving pain intensity | Count of | Dinama | Treatment policy | FAS | LR | J2R-MI |
| (NRS) reduction ≥50%<br>(yes/no) | subject | Binary | Hypothetical | FAS | LR | MMRM |

<sup>\*)</sup> Thresholds for meaningful within-subject change are presented in Table 2-6

#### 2.4.4 Exploratory endpoints

Exploratory endpoints are listed in section 1.1.3.4. All tests are tests of superiority of semaglutide s.c. 2.4 mg once-weekly to semaglutide placebo.

#### Analyses addressing the secondary estimand

The endpoints related to SF-36 addressing the secondary estimand will be analysed using the same imputation approach as used for the primary endpoints. The statistical model for continuous endpoints will be the same linear regression as for the primary endpoints (ANCOVA) with treatment as a factor and the baseline value of the endpoint as covariate.

#### Analyses addressing the additional estimand

The endpoints related to SF-36 addressing the additional estimand will be analysed using the same MMRM as described for the primary endpoints addressing the additional estimand with randomised treatment as a factor and the baseline value of the endpoint as covariate.

#### Other analyses

The endpoint change in 6 minutes walking distance from baseline to end of treatment will be summarised using descriptive statistics.

SAP NN9536-4578 SAP | 26 of 28

Statistical Analysis Plan

Date: 13 November 2023 Novo Nordisk
Trial ID: NN9536-4578

CONFIDENTIAL Version: 6.0

| CONFIDENTIAL | Version: 6.0 | Status: Final |

Table 2-8 Analysis and imputation methods to address the secondary and additional estimands for exploratory endpoints.

| Endpoint title | Unit | Endpoint Strategy | | Analysis set | Statistical<br>model | Imputation approach |
|---|---|---|---|---|---|---|
| Change in 6 minutes walking distance | Meters | Continuous | - | FAS | Descriptive statistics | - |
| Change in SF-36 role- | Score | Continuous | Treatment policy | FAS | ANCOVA | RD-MI |
| physical score | points | Continuous | Hypothetical | FAS | MMRM | - |
| Change in SF-36 general | Score | Cantina and | Treatment policy | FAS | ANCOVA | RD-MI |
| health score | points | Continuous | Hypothetical | FAS | MMRM | - |
| Change in SF-36 vitality | Score | a i | Treatment policy | FAS | ANCOVA | RD-MI |
| score | points | Continuous | Hypothetical | FAS | MMRM | - |
| Change in SF-36 social | Score | a i | Treatment policy | FAS | ANCOVA | RD-MI |
| functioning score | points | Continuous | Hypothetical | FAS | MMRM | - |
| Change in SF-36 role- | Score | a i | Treatment policy | FAS | ANCOVA | RD-MI |
| emotional score | points | Continuous | Hypothetical | FAS | MMRM | - |
| Change in SF-36 mental | Score | G .: | Treatment policy | FAS | ANCOVA | RD-MI |
| health score | points | Continuous | Hypothetical | FAS | MMRM | - |

### Analysis of safety endpoints

Adverse events will be defined as "treatment-emergent" (TEAE), if the onset of the event occurs in the on-treatment period. TEAEs and SAEs will be summarised by descriptive statistics, such as frequencies and rates. No formal statistical inference will be carried out based on the number of TEAEs and SAEs. All AEs will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA).

SAP NN9536-4578 SAP 27 of 28

Statistical Analysis Plan
Trial ID: NN9536-4578
EudraCT No: 2017-003436-36

Status: Final 

## 3 References

- 1. McEvoy BW. Missing data in clinical trials for weight management. J Biopharm Stat. 2016;26(1):30-6.
- 2. Carpenter JR, Roger JH, Kenward MG. Analysis of longitudinal trials with protocol deviation: a framework for relevant, accessible assumptions, and inference via multiple imputation. J Biopharm Stat. 2013;23(6):1352-71.
- 3. Sacks FM, Bray GA, Carey VJ, Smith SR, Ryan DH, Anton SD, et al. Comparison of weight-loss diets with different compositions of fat, protein, and carbohydrates. N Engl J Med. 2009;360(9):859-73
- 4. Bliddal H, Leeds AR, Stigsgaard L, Astrup A, Christensen R. Weight loss as treatment for knee osteoarthritis symptoms in obese patients: 1-year results from a randomised controlled trial. Ann Rheum Dis. 2011;70(10):1798-803.
- 5. Christensen R, Astrup A, Bliddal H. Weight loss: the treatment of choice for knee osteoarthritis? A randomized trial. Osteoarthritis Cartilage. 2005;13(1):20-7.
- 6. Bellamy. Comparison of transformed analogue and native numeric rating scaled patient responses to the WOMAC Index Internal Medicine Journal 2011;41(Suppl. s1):23.

SAP NN9536-4578 SAP 28 of 28





# Memo

To: NN9536-4578 Trial Squad

Copy: From: Pages: 1

November 22, 2023

## Post-hoc analysis for responder endpoint

Post DBL, for the responder endpoint of body weight reduction >= 20% at week 68, the model originally specified in the SAP for binary endpoints could not be fit as there were no responders in the placebo group. Hence a post-hoc analysis using Firth's approximation was performed using logistic regression with Firth's penalized likelihood.

Novo Nordisk A/S Biostatistics Vandtårnsvej 114 DK-2860 Søborg Denmark Telephone: +45 4444 8888 Direct dial: E-mail:

Internet:
www.novonordisk.com

Filenote Post-hoc analysis 1 of 1

# SAS dataset MedDRA terms for PROJECTs NN9536, EX9536 and NN9932 ReqNo: 2706 Print of SAS dataset named: NN9536\_EX9536\_NN9932\_v260 MedDRA version: 260


| | 396 congenital 1001033 | 1 genetic disorders 260 | 0 |
|---|---|---|---|
| | | Congenital, familial and genetic disorders 260 | ;0 |
| Rare events BROAD 10082036 decreased 10047938 White blood cell analyses 100188 | Haematology investigations (incl blood groups) 1002288 Neurological disorders | 1 Investigations 260 Congenital, tamilial and | .0 |
| | 299 congenital 1001033 | 1 genetic disorders 260 | 0 |
| Short stature homeobox Gene mutations and other Rare events NARROW 10082164 gene mutation 10083625 alterations NEC 100836 | abnormalities, gene<br>alterations and gene<br>324 variants 100103 | Congenital, familial and 1 genetic disorders 260 | 60 |
| Gap junction protein beta 2 Gene mutations and other | abnormalities, gene<br>alterations and gene | Congenital, familial and 1 genetic disorders 260 | 60 |
| Congenital nasal septum | Respiratory disorders | Congenital, tamilial and<br>1 genetic disorders 260 | i0 |
| Muscuroskeletar and Shprintzen-Goldberg connective tissue disorders | musculoskeletal and connective tissue disorders | Congenital, familial and genetic disorders 260 | |
| MUSCUUDSREHEIR AITO CONNECTIVE IBSUE disorders | musculoskeletal and connective tissue disorders | Congenital, familial and genetic disorders 260 | 60 |
| Alpha-thalassaemia-Haemoglobinopathies Rare events NARROW 10082291 intellectual deficit syndrome 10018903 congenital 100052 | system disorders | Congenital, familial and genetic disorders 260 | <del>-</del> |
| wuscuussemena anu<br>connective tissue disorders<br>of face, neck and jaw | Musculoskeletal and connective tissue disorders congenital 1001033 | Congenital, familial and genetic disorders 260 | ;0 |
| X-linked intellectual Gene mutations and other Rare events NARROW 10082377 disability, Siderius type 10083625 alterations NEC 100836 | | Congenital, familial and genetic disorders 260 | ;O |
| | | Congenital, familial and genetic disorders 260 | ;0 |
| Rare events NARROW 10082379 syndrome 10027671 congenital NEC 100146 | | Congenital, tamilial and<br>1 genetic disorders 260 | 0 |
| Rare events NARROW 10082380 Aberrant aortic arch 10018717 congenital 100075 | | Congenital, tamilial and<br>1 genetic disorders 260 | i0 |
| Non-site specific cartilage Rare events NARROW 10082381 SADDAN syndrome 10029510 disorders congenital 100286 | musculoskeletal and connective tissue disorders congenital 1001033 | Congenital, familial and genetic disorders 260 | ;0 |
| | abnormalities, gene<br>alterations and gene<br>324 variants 1001033 | Congenital, familial and genetic disorders 260 | ;0 |
| Rare events NARROW 10082393 Hyperpipecolic acidaemia 10021602 metabolism 100277 | Metabolic and nutritional<br>424 disorders congenital 1001033 | Congenital, tamilial and<br>1 genetic disorders 260 | i0 |
| Rare events NARROW 10082398 1p36 deletion syndrome 10029513 congenital NEC 100285 | musculoskeletar and connective tissue disorders congenital 1001033 musculoskeletar and | Congenital, familial and genetic disorders 260 | ;0 |
| | connective tissue disorders<br>396 congenital 1001033 | Congenital, familial and<br>1 genetic disorders 260 | ;0 |
| | | Congenital, tamilial and genetic disorders 260 | .0 |
| Rare events NARROW 10082546 occlusion 10003153 congenital 100075 | Cardiac and vascular 510 disorders congenital 1001033 | Congenital, ramiliar and<br>1 genetic disorders 260 | 0 |
| Plasminogen activator Coagulation disorders | system disorders | Congenital, familial and 1 genetic disorders 260 Congenital, familial and | 0 |
| Rare events NARROW 10082603 deficiency 1000140 derican disorders 100140 deficiency 1000140 def | 599 congenital 1001033 | 1 genetic disorders 260 | .0 |
| | | Congenital, familial and genetic disorders 260 | ;0 |
| Rare events NARROW 10082605 Uterine cervix canal atresia 10016416 disorders congenital 100386 | Reproductive tract and breast disorders congenital 1001033 | Congenital, ramilial and genetic disorders 260 | .0 |
| brain iron accumulation Central nervous system | Neurological disorders 299 congenital 1001033 | Congenital, familial and genetic disorders 260 | 0 |
| Apolipoprotein E e4 gene | abnormalities, gene<br>alterations and gene<br>324 variants 1001033 | Congenital, familial and<br>1 genetic disorders 260 | ;0 |
| Rare events NARROW 10082665 Double inlet left ventricle 10028177 abnormalities congenital 100075 | | Congenital, tamilial and<br>1 genetic disorders 260 | 10 |
| Congenital Dilateral Cerebral disorders | Neurological disorders<br>299 congenital 1001033 | Congenital, tamilial and<br>1 genetic disorders 260 | ·0 |


# Meaningful Within-Patient Change in Patient-Reported Outcome Measures of Pain and Physical Functioning in Patients With Obesity and Osteoarthritis of the Knee

Psychometric Analysis Plan for NN9536-4578 Final (Version 1.0)

### 24 January 2022

Prepared for

Novo Nordisk A/S

Prepared by



Project No. 0306398.000

### **APPROVALS**

Meaningful Within-Patient Change in Patient-Reported Outcome Measures of Pain and Physical Functioning in Patients With Obesity and Osteoarthritis of the Knee: Final Psychometric Analysis Plan; Version 1.0; 24 January 2022

### **PRIMARY AUTHOR**

Your signature below indicates that this document is accurate and complete.

### **PRIMARY APPROVERS**

Your signature below indicates that this document is accurate and complete.



### **DOCUMENT VERSION HISTORY**

| Date | Description |
|-------------|---------------------------------|
| 14 Dec 2021 | Draft delivered to Novo Nordisk |
| 24 Jan 2022 | Final delivered to Novo Nordisk |

## **TABLE OF CONTENTS**

| 1 | INTRODUCTION | 7 |
|------------|-----------------------------------------------------------|-----|
| 2 | ANALYSIS OBJECTIVES | 7 |
| 3 | DATA FOR THE PLANNED ANALYSES | 7 |
| 3.1 | Data Set Description and Structure | |
| 3.2 | Data Security | |
| 4 | SOFTWARE TOOLS AND ANALYSIS PACKAGES | 8 |
| 5 | DATA SOURCE | 8 |
| 5.1 | Study Design | 8 |
| | 5.1.1 Key Eligibility Criteria | 9 |
| 5.2 | Analysis Data | 10 |
| 6 | MEASURES | 11 |
| 6.1 | Western Ontario and McMaster Universities Arthritis Index | 11 |
| 6.2 | SF-36 Health Survey, Acute Version 2 | |
| 6.3 | Patient Global Impression Items for Pain | |
| 6.4 | Patient Global Impression Items for Physical Functioning | |
| 6.5 | Body Weight | |
| 7 | PROPOSED ANALYSES | |
| 7.1 | Analysis Conventions | |
| 7.2<br>7.3 | Missing Data | |
| 7.3<br>7.4 | Descriptive Statistics Evaluation of Anchors | |
| 7.5 | Meaningful Within-Patient Change | |
| | 7.5.1 Anchor-Based Methods | |
| | 7.5.2 Distribution-Based Methods | |
| 8 | REFERENCES | |
| • | | |
| APP | ENDIX A. TABLE SHELLS | A-1 |
| APP | ENDIX B. FIGURE TEMPLATES | B-1 |

### **TABLES**

| Table 1. | Schedule of Key Timepoints Relevant to Psychometric Analyses 11 |
|---|---|
| Table 4. | SF-36 Health Survey, Acute Version 2: Physical Functioning Subscale 13 |
| Table A-1. | Patient Characteristics (Baseline Values)A-2 |
| Table A-2. | Descriptive Statistics for WOMAC Pain, WOMAC Physical Functioning, and SF-36v2 Physical Functioning ScoresA-3 |
| Table A-3. | Response Frequency (%) Distributions for Supporting MeasuresA-4 |
| Table A-4. | Descriptive Statistics of Supporting MeasuresA-5 |
| Table A-5. | Correlations Between WOMAC Pain, WOMAC Physical Functioning, and SF-36v2 Physical Functioning Scores and Supporting MeasuresA-6 |
| Table A-6. | Descriptive Statistics of the Changes in WOMAC and SF-36v2 Subscale Scores by Changes in Candidate Anchor MeasuresA-7 |
| Table A-7. | Frequencies and Percentages of Crosstabulation Between Changes in PGI-S and PGI-C Items at Week 68 |
| Table A-8. | Change in WOMAC Pain in Patients Who Achieved a 1-Point PGI-S for Pain Improvement From Baseline to Week 68 |
| Table A-9. | Change in WOMAC Pain in Patients Who Achieved a 2-Point PGI-S for Pain Improvement From Baseline to Week 68 |
| Table A-10. | Change in WOMAC and SF-36v2 Physical Functioning in Patients Who Achieved a 1-Point PGI-S for PF Improvement From Baseline to Week 68 |
| Table A-11. | Change in WOMAC and SF-36v2 Physical Functioning in Patients Who Achieved a 2-Point PGI-S for PF Improvement From Baseline to Week 68 |
| Table A-12. | Interpretation of Change: Distribution-Based Method |

## **FIGURES**

| Figure B-1. | Empirical Cumulative Distribution Function Plot of Change in Target Clinical Outcome Assessment Score, by Change in Anchor MeasureB- |
|---|---|
| Figure B-2. | Probability Density Function Plot of Change in Target Clinical Outcome Assessment Score, by Anchor Measure |

### **ABBREVIATIONS**

| Abbreviation | Term |
|--------------|-----------------------------------------------------------|
| 6MWD | 6-minute walking distance |
| ACR | American College of Rheumatology |
| ADaM | Analysis Data Model |
| BMI | body mass index |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | confidence interval |
| COA | clinical outcome assessment |
| eCDF | empirical cumulative distribution function |
| EOT | end of treatment |
| FDA | Food and Drug Administration |
| max | maximum |
| min | minimum |
| MCS | Mental Component Summary |
| MWPC | meaningful within-patient change |
| Novo Nordisk | Novo Nordisk A/S |
| NRS | numeric rating scale |
| OA | osteoarthritis |
| PCS | Physical Component Summary |
| PDF | probability density function |
| PF | Physical Functioning |
| PGI-C | Patient Global Impression of Change |
| PGI-S | Patient Global Impression of Status |
| PRO | patient-reported outcome |
| s.c. | subcutaneous |
| SD | standard deviation |
| SF-36v2 | SF-36 Health Survey, Acute Version 2.0 |
| WOMAC | Western Ontario and McMaster Universities Arthritis Index |

### 1 INTRODUCTION

Novo Nordisk A/S (Novo Nordisk) is conducting a phase 3b trial (NN9536-4578) of semaglutide in patients with obesity and knee osteoarthritis (OA). Two patient-reported outcome (PRO) measures—the Western Ontario and McMaster Universities Arthritis Index (WOMAC) and the SF-36 Health Survey, Acute Version 2 (SF-36v2)—have been included in this trial to support key endpoints. Specifically, changes in the WOMAC Pain subscale score will be evaluated alongside changes in body weight as primary endpoints; changes in the WOMAC and SF-36v2 Physical Functioning (PF) subscale scores will be evaluated as confirmatory secondary endpoints.

In preparation for a submission to the Food and Drug Administration (FDA) in early 2020, collaborated with Novo Nordisk on the development of a briefing document supporting use of the WOMAC and SF-36v2 in NN9536-4578. The FDA has since provided written feedback, including recommendations regarding the assessment of meaningful change on the WOMAC Pain and PF subscales and on the SF-36v2 PF subscale.

### 2 ANALYSIS OBJECTIVES

The analyses described in this psychometric analysis plan are intended to address the FDA's feedback regarding estimation and support of meaningful within-patient change (MWPC) thresholds for the WOMAC Pain and PF subscales and on the SF-36v2 PF subscale, using data from patients in NN9536-4578. The analysis methods have been planned in accordance with the recommendations outlined in FDA guidance documents pertaining to PRO measures and other types of clinical outcome assessments (COAs) (FDA, 2009; 2018a; 2018b).

### 3 DATA FOR THE PLANNED ANALYSES

This psychometric evaluation will use data from NN9536-4578, a phase 3b trial designed to assess the efficacy and safety of semaglutide subcutaneous (s.c.) 2.4 mg administered once weekly in patients with obesity and knee OA.

### 3.1 Data Set Description and Structure

will be responsible for creating the analysis data sets based on fully deidentified Analysis Data Model (ADaM) trial data sets provided by Novo Nordisk that are compliant with the Clinical Data Interchange Standards Consortium (CDISC) guidelines and are provided as SAS data sets or in SAS transport format.

anticipates that the analysis data sets will include the following (at a minimum): basic demographics; scores for the WOMAC Pain and PF subscales and the SF-36v2 PF subscale (visit scores and changes from baseline, as well as raw and transformed scores where applicable); responses to global items assessing patients' perceptions of their current status and changes (from baseline) in their knee pain and physical functioning; and percent changes in body weight.

Novo Nordisk will be responsible for reviewing and approving descriptive statistics produced by based on the derived analysis data. Upon approval of the descriptive statistics, will complete the remaining planned analyses described in this psychometric analysis plan.

### 3.2 Data Security

The deidentified data set will be stored in a secure location (accessible only to authorized members of the project team) on a qualified server located on the campus of Specifically, the data will reside on a Federal Information Processing Standard–Low Certified and Accredited Network, which is compliant with all required controls, including physical and logical security, environmental conditioning, and automatic monitoring.

### 4 SOFTWARE TOOLS AND ANALYSIS PACKAGES

Following standard practice for psychometric evaluations, most of the planned analyses will be performed using SAS version 9.4 in a Linux-based environment (Cary, NC: SAS Institute, Inc.; 2013). Other commercially available psychometric analysis packages will be used where appropriate.

### 5 DATA SOURCE

### 5.1 Study Design

NN9536-4578 is a phase 3b, randomized, double-blinded, placebo-controlled, multicenter clinical trial designed to investigate the effects of semaglutide s.c. 2.4 mg, administered once weekly, in adults with moderate OA of one or both knees, pain due to knee OA, and obesity (body mass index [BMI]  $\geq$  30.0 kg/m²). Trial participants will be randomized in a 2:1 manner to receive either semaglutide s.c. 2.4 mg or semaglutide placebo once weekly as an adjunct to a reduced-calorie diet and increased physical activity. Approximately 420 patients will be screened to achieve 375 participants randomly assigned to the trial product.

The total trial duration for an individual participant will be approximately 76 weeks. The trial includes a screening period of approximately 1 week followed by randomization. Dose escalation of semaglutide/semaglutide placebo will take place every 4 weeks during the first 16 weeks after randomization. Following dose escalation, visits are scheduled every eighth week until the end of treatment (EOT) at week 68. The follow-up period is 7 weeks after EOT.

The primary endpoints include change in WOMAC Pain subscale scores and percentage change in body weight from baseline/week 0 to EOT/week 68. The confirmatory secondary endpoints include the proportions of patients losing at least 5% and 10% of their baseline body weight at week 68 and changes in WOMAC PF and SF-36 PF subscale scores from baseline to week 68. Additional secondary endpoints include change from baseline to week 68 in waist circumference; WOMAC Stiffness and Total scores; SF-36v2 Bodily Pain subscale, Physical Component Summary, and Mental Component Summary scores; use of analgesics; and pain intensity. Changes from baseline to week 68 in additional SF-36v2 scores and 6-minute walking distance (6MWD) will be evaluated as exploratory endpoints. All trial endpoints are detailed in Section 3.2 of Protocol NN9536-4578 (Version 3.0, Final, 21 April 2021).

### 5.1.1 Key Eligibility Criteria

This section presents key eligibility criteria used to recruit participants for the trial.

Additional details can be found in Protocol NN9536-4578 (Version 3.0, Final, 21 April 2021).

Key inclusion criteria are as follows:

- Male or female, aged ≥ 18 years at the time of signing informed consent
- BMI  $\geq$  30.0 kg/m<sup>2</sup>
- Clinical diagnosis of knee OA (American College of Rheumatology [ACR] criteria) with moderate radiographic changes (Kellgren-Lawrence grades 2 or 3 as per central reading) in target knee. Target knee joint is defined as most symptomatic knee at screening. If pain is equal in both knees, the target knee joint will be in the most dominant leg
- Pain due to knee OA, with randomization criteria:
  - 1. A score of at least 40 on the WOMAC Pain subscale
  - For patients taking analgesics, attend randomization visit after 72-hour washout period (rescue medication with acetaminophen allowed until 24 hours before visit)

Key exclusion criteria are as follows:

- Joint replacement in target knee
- · Arthroscopy or injections into target knee within last 3 months prior to enrollment
- Any other joint disease in the target knee

### 5.2 Analysis Data

The psychometric analyses will use NN9536-4578 data from the screening period (visit 1), baseline/week 0 (visit 2), week 20 (visit 7), and week 68 (visit 13). Table 1 presents the schedule of events relevant to the planned analyses. Additionally, the psychometric analysis sample will only use data from patients in the full analysis set of the trial who have a nonmissing score for at least 1 target endpoint (WOMAC Pain, WOMAC PF, or SF-36v2 PF) at baseline.

Consistent with the FDA's recommendations, receipt of a preliminary data set is expected after approximately 100 patients have completed the trial (projected by Novo Nordisk to occur in July 2023). Most of the planned analyses (including descriptive statistics, correlational analyses, descriptive anchor-based estimation, and distribution-based estimation) will be conducted using the preliminary data set, and the results will be supplemented by conducting the same analyses and the remaining analyses (i.e., graphical displays and sensitivity analyses) using the final (full) data set. The estimation results from the final data set, specifically those based on the Patient Global Impression of Status (PGI-S) Pain and PF items, will provide the primary MWPC thresholds to be used by Novo Nordisk in support of the clinical efficacy analyses; however, ranges of plausible thresholds for the WOMAC Pain, WOMAC PF, and SF-36v2 PF scores will be provided to the FDA before unblinding.

Table 1. Schedule of Key Timepoints Relevant to Psychometric Analyses

| | Baseline<br>(week 0, randomization) | Week 20<br>(treatment period) | EOT<br>(week 68) |
|---|---|---|---|
| Information | Visit 2 | Visit 7 | Visit 13 |
| Patient information | | | |
| Demography | Χa | | |
| Height | Χa | | |
| Target measures | | | |
| WOMAC | X | X | X |
| SF-36v2 | X | X | X |
| PGI-S for Pain | X | X | X |
| PGI-C for Pain | | Х | X |
| PGI-S for Physical Function | X | Х | X |
| PGI-C for Physical Function | | Х | X |
| Body weight | X | Х | Х |

EOT = end of treatment; PGI-C = Patient Global Impression of Change; PGI-S = Patient Global Impression of Status; SF-36v2 = SF-36 Health Survey, Acute Version 2; WOMAC = Western Ontario and McMaster Universities Arthritis Index

### 6 MEASURES

### 6.1 Western Ontario and McMaster Universities Arthritis Index

The WOMAC is a disease-specific PRO measure designed to assess changes in symptoms and lower extremity functioning associated with treatment in patients with OA of the hip and knee (Bellamy et al., 1988). The WOMAC comprises 24 items across 3 subscales: Pain (5 items), PF (17 items), and Stiffness (2 items); a Total score can also be computed. Version 3.1 of the WOMAC will be administered in NN9536-4578. It includes numeric rating scale (NRS) responses ranging from no symptom/difficulty (0) to extreme symptom/difficulty (10) and uses a 24-hour recall period. The items comprising the Pain and PF subscales are shown in Table 2 and Table 3, respectively. For each of them, corresponding raw item scores are summed and transformed a standardized 0 (best) to 100 (worst) score range.

<sup>&</sup>lt;sup>a</sup> Baseline values collected at screening (visit 1).



In NN9536-4578, the WOMAC will be completed using an electronic device during all 12 clinical visits from baseline/randomization (week 0) to EOT (week 68). The planned analyses will use WOMAC data collected at baseline (week 0), week 20, and week 68.

### 6.2 SF-36 Health Survey, Acute Version 2

The SF-36/SF-36v2 (Ware and Sherbourne, 1992) is a widely used, generic self-report measure of perceived health status. The SF-36v2 contains 36 items that are scored as 8 multiple-item subscales addressing the following concepts: physical functioning, role limitations due to physical health problems, bodily pain, social functioning, general mental health, role limitations due to emotional problems, vitality, and general health perceptions. There are also 2 summary scores, a Physical Component Summary (PCS) score and a Mental Component Summary (MCS) score. Each SF-36v2 component and subscale is scored from 0 to 100, with higher scores indicating better functioning. The acute form of this measure, planned for inclusion in NN9536-4578, uses a 1-week recall period.

The 10 items comprising the SF-36v2 PF subscale are shown in Table 4.

Table 4. SF-36 Health Survey, Acute Version 2: Physical Functioning Subscale

| dui | e following questions are about activities you might do<br>ring a typical day. Does <u>your health now limit you</u> in<br>se activities? If so, how much? | Yes,<br>limited<br>a lot<br>▼ | Yes,<br>limited<br>a little<br>▼ | No, not<br>limited<br>at all<br>▼ |
|---|---|---|---|---|
| а | <u>Vigorous activities</u> , such as running, lifting heavy objects, participating in strenuous sports | | | |
| b | <u>Moderate activities</u> , such as moving a table, pushing a vacuum cleaner, bowling, or playing golf | | | |
| С | Lifting or carrying groceries | | | |
| d | Climbing several flights of stairs | | | |
| е | Climbing one flight of stairs | | | |
| f | Bending, kneeling, or stooping | | | |
| g | Walking more than a mile | | | |
| h | Walking several hundred yards | | | |
| i | Walking one hundred yards | | | |
| j | Bathing or dressing yourself | | | |

In NN9536-4578, the SF-36v2 form will be completed using an electronic device during the following clinic visits: 2 (week 0), 4 (week 8), 7 (week 20), 9 (week 36), 11 (week 52), and 13 (week 68). The current analyses will use SF-36v2 data collected at baseline (week 0), week 20, and week 68.

### 6.3 Patient Global Impression Items for Pain

A single-item PGI-S for Pain will be administered in NN9536-4578 at baseline (week 0) and weeks 20, 52, and 68. The PGI-S for Pain asks patients to rate their current knee pain ("How would you rate the severity of your knee pain currently?"), using a 4-point ordinal scale (none, mild, moderate, and severe). The current analyses will use PGI-S for Pain responses collected at baseline, week 20, and week 68.

At week 20, week 52, and week 68, a single-item Patient Global Impression of Change (PGI-C) for Pain will also be administered. The PGI-C for Pain asks patients to rate any changes in their knee pain since baseline ("Compared to the beginning of the study, how would you rate your knee pain currently?") using a 7-point scale (much better, moderately better, a little better, no difference, a little worse, moderately worse, or much worse). The current analyses will use PGI-C for Pain responses collected at week 20 and week 68.

### 6.4 Patient Global Impression Items for Physical Functioning

A single-item PGI-S for PF will be administered in NN9536-4578 at baseline (week 0), as well as weeks 20, 52, and 68. The PGI-S for PF asks patients to rate their current functioning ("How would you rate your physical functioning [mobility and ability to do physical activities] currently?") using a 5-point ordinal scale (poor, fair, good, very good, and excellent). The current analyses will use PGI-S for PF responses collected at baseline (week 0), week 20, and week 68.

At week 20, week 52, and week 68, a single-item PGI-C for PF will also be administered. The PGI-C for PF asks patients to rate any changes since baseline in their functioning ("Compared to the beginning of the study, how would you rate your physical functioning [mobility and ability to do physical activities] currently?") using a 7-point scale (much better, moderately better, a little better, no difference, a little worse, moderately worse, or much worse). The current analyses will use PGI-C for PF responses collected at week 20 and week 68.

### 6.5 Body Weight

In NN9536-4578, body weight will be measured at the following clinic visits: 1 (screening), 2 (baseline/week 0), 4 (week 8), 7 (week 20), 9 (week 36), 11 (week 52), and 13 (week 68). The current analyses will use the data collected at baseline (week 0), week 20, and week 68.

### 7 PROPOSED ANALYSES

### 7.1 Analysis Conventions

Analyses will be conducted without regard to treatment assignment. Observed data from patients who discontinue the trial will be also included. The scoring of the relevant measures will be performed by Novo Nordisk.

For analyses related to interpretation of change, if very few patients ( $n \le 5$ ) are in a category defined by the anchor measure, adjacent categories (e.g., "moderately worse" and "much worse" for a PGI-C item) may be collapsed. Results will be reported using the uncollapsed and collapsed (if applicable) categories. For other planned analyses beyond descriptive statistics, a footnote and "—" will denote cases in which statistical results are not reported due to small sample sizes (i.e.,  $n \le 5$ ).

Appendix A presents the table templates and Appendix B presents the figure templates for the planned analyses.

### 7.2 Missing Data

Missing scores for the WOMAC, SF-36v2, PGI-S, and PGI-C will not be imputed (e.g., no use of last observation outside scheduled window carried forward). Other measures used in the evaluation will be scored according to Novo Nordisk's data management plans for scoring.

### 7.3 Descriptive Statistics

Standard descriptive statistics will be presented to summarize sample characteristics (Table A-1).

For the WOMAC Pain and PF scores, as well as the SF-36v2 PF scores, the following descriptive statistics will be tabulated:

- Standard descriptive statistics (e.g., means, standard deviations [SDs], floor [worst score] and ceiling [best score] percentages, missingness) of the scores at baseline (week 0), week 20, and week 68 (Table A-2)
- Standard descriptive statistics (e.g., means, SDs, missingness) for the change scores from baseline (week 0) to week 20 and week 68 (Table A-2)

The descriptive statistics of the potential anchor measures and other supporting measures are as follows:

 Response frequencies of PGI-S items at baseline, week 20, and week 68; response frequencies of PGI-C items and weight change categories at week 20 and week 68 (Table A-3) Standard descriptive statistics (e.g., means, SDs, missingness) of PGI-S items, PGI-C items, and body weight at baseline (PGI-S and body weight only), week 20, and week 68, as well as the changes in the PGI-S items and percentage change in body weight from baseline to week 20 and week 68 (Table A-4)

### 7.4 Evaluation of Anchors

To support the selection of appropriate anchors for the estimation of MWPC thresholds for the WOMAC and SF-36v2 subscale scores, analyses will be conducted to evaluate the scores' ability to detect change in patients whose clinical status has changed.

Longitudinal correlations will be computed between the changes in the WOMAC Pain, WOMAC PF, and SF-36v2 PF subscales and the candidate anchor measures from baseline to week 20 and week 68 (Table A-5).

It is recommended to select an anchor measure with responsiveness correlation magnitude greater than 0.30 according to Revicki and colleagues (2008) or 0.371 according to Hays et al. (2005). Stronger correlations between the target COA and the anchor measures generally help to reduce the anchor-based estimation confidence intervals (Qin et al., 2017).

Descriptive statistics of the changes in WOMAC Pain, WOMAC PF, and SF-36v2 PF subscale scores by the changes in candidate anchor measures (i.e., changes in PGI-S items, PGI-C item responses, and percent changes in body weight) will be reviewed (Table A-6). The size and direction of the group mean and median changes in WOMAC and SF-36v2 scores should follow a predictable pattern; that is, the greater improvement or worsening in the target PRO scores should be achieved by patients who show greater levels of improvement or worsening on appropriate anchor measures, respectively.

### 7.5 Meaningful Within-Patient Change

The anchor-based method (using the PGI-S and PGI-C items, as well as percent change in body weight) and a supportive, distribution-based method (half-SD at baseline) will be used to establish MWPC thresholds for the target WOMAC and SF-36v2 subscale scores.

### 7.5.1 Anchor-Based Methods

Anchor-based methods use external criteria (e.g., global impression measures or established and validated measures) to estimate thresholds for changes in the target instrument that are clinically relevant.

The PGI-S and PGI-C items, as well as percent change in body weight, are candidate anchor measures for the MWPC thresholds for improvement on the target WOMAC and SF-36v2

subscale scores. To be considered an appropriate anchor, the responsiveness correlation between the candidate anchor and the target PRO measure (WOMAC or SF-36v2 subscale score) must be at least 0.371 and descriptive mean changes must follow the anticipated pattern. To further support the meaningfulness of the anchor levels, a crosstabulation between the change in each PGI-S item and the corresponding PGI-C item will be reported (Table A-7). If a PGI-S item is confirmed as an appropriate anchor, a 1-point improvement in PGI-S will be considered the primary anchor for the corresponding target PRO score, and the MWPC threshold of the change in corresponding target PRO score (i.e., responder definition) will be estimated as the mean change from baseline to week 68 (bolded rows in Table A-6).

The anchor-based estimates for MWPC thresholds (mean changes from baseline to week 68 in the target PRO score) will be also considered as supportive at the following anchor levels:

- PGI-C for Pain category "moderately better" at week 68 for the WOMAC Pain subscale score
- PGI-C for PF category "moderately better" at week 68 for the WOMAC PF and SF-36v2 PF subscale scores
- Weight loss between 5% and 10% of baseline body weight at week 68 for all 3 target PRO scores

Additional supportive anchor-based estimates for MWPC thresholds will be computed using the same anchor levels and change from baseline to week 20 (Table A-6).

As sensitivity analyses (Table A-8-Table A-11), descriptive statistics of the changes in the target WOMAC and SF-36v2 subscale scores by baseline PGI-S categories will be reported in patients who achieved a 1-point PGI-S improvement, as well as those who achieved a 2-point PGI-S improvement from baseline to week 68. The sensitivity analyses will be conducted only for the final data set.

### 7.5.1.1 Graphical Displays

To provide graphical support for the anchor measures, empirical cumulative distribution function (eCDF) and probability density function (PDF) plots will be produced for the changes in target WOMAC and SF-36v2 subscale scores by the changes in anchor measures deemed appropriate from baseline to week 68 (Figure B-1 and Figure B-2). The eCDF curves help elucidate the impact of different threshold choices. The spread, height, and separation of the PDF curves offer an intuitive understanding of the discriminating ability of the different levels of the anchor variable. Ideally, curves in both plots should be distinct and ordered from worst (negative changes) to best (positive changes) along the horizontal axis. The graphic displays will be generated only for the baseline to week 68 changes in the final data set.

### 7.5.2 Distribution-Based Methods

A supportive, distribution-based method will also be applied to explore thresholds for MWPC (Table A-12). The half-SDs of baseline WOMAC and SF-36v2 subscale scores, which correspond to moderate effect sizes (Cohen, 1992), will be computed.

### 8 REFERENCES

- Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988;15(12):1833-40.
- Cohen J. A power primer. Psych Bull. 1992;112(1):155-9. doi:10.1037//0033-2909.112.1.155.
- FDA. Food and Drug Administration. Guidance for industry: patient-reported outcome measures: use in medical product development to support labeling claims. 2009. <a href="https://www.fda.gov/downloads/Drugs/Guidances/ucm193282.pdf">https://www.fda.gov/downloads/Drugs/Guidances/ucm193282.pdf</a>. Accessed 10 October 2021.
- FDA. Food and Drug Administration. Patient-focused drug development (PFDD) guidance: methods to identify what is important to patients & select, develop or modify fit-for-purpose clinical outcomes assessments. Guidance 3 discussion document. October 15-16, 2018a. <a href="https://www.fda.gov/media/116277/download">https://www.fda.gov/media/116277/download</a>. Accessed 24 November 2021.
- FDA. Food and Drug Administration. Patient-focused drug development (PFDD) guidance: methods to identify what is important to patients & select, develop or modify fit-for-purpose clinical outcomes assessments. Attachment to guidance 3 discussion document appendices. October 15-16, 2018b. <a href="https://www.fda.gov/media/116281/download">https://www.fda.gov/media/116281/download</a>. Accessed 24 November 2021.
- Hays RD, Farivar SS, Liu H. Approaches and recommendations for estimating minimally important differences for health-related quality of life measures. J Chron Obstruct Pulmon Dis. 2005 Mar;2(1):63-7. doi:10.1081/copd-200050663.
- Qin S, Coles T, Nelson L, Williams V, Williams N, McLeod L. What impacts the stability of anchor-based responder definitions? Podium presentation at the International Society for Quality of Life Research 24th Annual Conference; 18-21 October 2017. Philadelphia, PA.

Revicki D, Hays R, Cella D, Sloan J. Recommended methods for determining responsiveness and minimally important differences for patient-reported outcomes. J Clin Epidemiol. 2008 Feb;61(2):102-9. doi:10.1016/j.jclinepi.2007.03.012.

Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992;30(6):473-83.

# Appendix A. Table Shells

Table A-1. Patient Characteristics (Baseline Values)

| | · |
|---|---|
| Patient characteristic | Overall<br>(N = xxx) |
| Age (years), mean (SD), n (%) | xx.x (xx.xx), xx (xx.x) |
| Median, min-max | XX.X, XX.X-XX.X |
| Sex, n (%) | ann, ann ann |
| Male | xx (xx.x) |
| Female | xx (xx.x) |
| Height (meters), mean (SD), n (%) | xx.x (xx.xx), xx (xx.x) |
| Median, min-max | XX.X, XX.X-XX.X |
| Weight (lb), mean (SD), n (%) | xx.x (xx.xx), xx (xx.x) |
| Median, min-max | XX.X, XX.X-XX.X |
| · | · |
| Weight (kg), mean (SD), n (%) Median, min-max | xx.x (xx.xx), xx (xx.x) |
| · | XX.X, XX.X-XX.X |
| BMI, mean (SD), n (%) Median, min-max | xx.x (xx.xx), xx (xx.x) |
| · | XX.X, XX.X-XX.X |
| Race, n (%) | and formal |
| White | xx (xx.x) |
| Black or African American | xx (xx.x) |
| Asian American | xx (xx.x) |
| Native American, American Indian, or Alaska<br>Native | xx (xx.x) |
| Native Hawaiian or Pacific Islander | xx (xx.x) |
| Another race | xx (xx.x) |
| Ethnicity, n (%) | |
| Hispanic, Latin American, or Latinx | xx (xx.x) |
| To be determined | |

BMI = body mass index; max = maximum; min = minimum; SD = standard deviation.

Table A-2. Descriptive Statistics for WOMAC Pain, WOMAC Physical Functioning, and SF-36v2 Physical Functioning Scores

| Score/timepoint | n | Mean (SD) | Median | Observed<br>min, max | Score<br>max (%)/<br>min (%) | Missing n<br>(%) |
|---|---|---|---|---|---|---|
| WOMAC Pain | | | | | | |
| Baseline | XX | xx.x (x.xx) | xx.x | xx, xx | xx.x/xx.x | xx (xx.x) |
| Week 20 | XX | xx.x (x.xx) | xx.x | xx, xx | xx.x/xx.x | xx (xx.x) |
| Week 68 | XX | xx.x (x.xx) | xx.x | xx, xx | xx.x/xx.x | xx (xx.x) |
| Change from baseline to week 20 | xx | xx.x (x.xx) | xx.x | xx, xx | - | xx (xx.x) |
| Change from baseline to week 68 | xx | xx.x (x.xx) | xx.x | xx, xx | - | xx (xx.x) |
| WOMAC PF | | | | | | |
| Baseline | XX | xx.x (x.xx) | xx.x | xx, xx | xx.x/xx.x | xx (xx.x) |
| Week 20 | XX | xx.x (x.xx) | xx.x | xx, xx | xx.x/xx.x | xx (xx.x) |
| Week 68 | XX | xx.x (x.xx) | xx.x | xx, xx | xx.x/xx.x | xx (xx.x) |
| Change from baseline to week 20 | XX | xx.x (x.xx) | xx.x | xx, xx | - | xx (xx.x) |
| Change from baseline to week 68 | xx | xx.x (x.xx) | xx.x | xx, xx | - | xx (xx.x) |
| SF-36v2 PF | | | | | | |
| Baseline | XX | xx.x (x.xx) | xx.x | xx, xx | xx.x/xx.x | xx (xx.x) |
| Week 20 | XX | xx.x (x.xx) | xx.x | xx, xx | xx.x/xx.x | xx (xx.x) |
| Week 68 | XX | xx.x (x.xx) | xx.x | xx, xx | xx.x/xx.x | xx (xx.x) |
| Change from baseline to week 20 | xx | xx.x (x.xx) | xx.x | xx, xx | - | xx (xx.x) |
| Change from baseline to week 68 | XX | xx.x (x.xx) | xx.x | xx, xx | - | xx (xx.x) |

max = maximum; min = minimum; PF = Physical Functioning; SD = standard deviation; SF-36v2 = SF-36 Health Survey, Acute Version 2.0; WOMAC = Western Ontario and McMaster Universities Arthritis Index.
Table A-3. Response Frequency (%) Distributions for Supporting Measures

| | | - | |
|---|---|---|---|
| Score | Baseline<br>(N = xxx) | Week 20<br>(N = xxx) | Week 68<br>(N = xxx) |
| PGI-S for Pain | | | |
| None | xx (x.x) | xx (x.x) | xx (x.x) |
| Mild | xx (x.x) | xx (x.x) | xx (x.x) |
| Moderate | xx (x.x) | xx (x.x) | xx (x.x) |
| Severe | xx (x.x) | xx (x.x) | xx (x.x) |
| PGI-C for Pain | | | |
| Much better | - | xx (x.x) | xx (x.x) |
| Moderately better | - | xx (x.x) | xx (x.x) |
| A little better | - | xx (x.x) | xx (x.x) |
| No difference | - | xx (x.x) | xx (x.x) |
| A little worse | - | xx (x.x) | xx (x.x) |
| Moderately worse | - | xx (x.x) | xx (x.x) |
| Much worse | - | xx (x.x) | xx (x.x) |
| PGI-S for PF | | | |
| Poor | xx (x.x) | xx (x.x) | xx (x.x) |
| Fair | xx (x.x) | xx (x.x) | xx (x.x) |
| Good | xx (x.x) | xx (x.x) | xx (x.x) |
| Very good | xx (x.x) | xx (x.x) | xx (x.x) |
| Excellent | xx (x.x) | xx (x.x) | xx (x.x) |
| PGI-C for PF | | | |
| Much better | - | xx (x.x) | xx (x.x) |
| Moderately better | - | xx (x.x) | xx (x.x) |
| A little better | - | xx (x.x) | xx (x.x) |
| No difference | - | xx (x.x) | xx (x.x) |
| A little worse | - | xx (x.x) | xx (x.x) |
| Moderately worse | - | xx (x.x) | xx (x.x) |
| Much worse | - | xx (x.x) | xx (x.x) |
| Percent weight change (reduction) | | | |
| < 5% | | xx (x.x) | xx (x.x) |
| 5 to 10% | | xx (x.x) | xx (x.x) |
| > 10% | | xx (x.x) | xx (x.x) |

PGI-C = Patient Global Impression of Change; PGI-S = Patient Global Impression of Status; PF = Physical Functioning.

Table A-4. Descriptive Statistics of Supporting Measures

| | | | | • | |
|---|---|---|---|---|---|
| Score/timepoint | n | Mean (SD) | Median | Observed<br>min, max | Missing<br>(%) |
| PGI-S for Pain | | | | | |
| Baseline | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| Week 20 | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| Week 68 | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| Change from baseline to week 20 | XX | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| Change from baseline to week 68 | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| PGI-S for PF | | | | | |
| Baseline | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| Week 20 | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| Week 68 | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| Change from baseline to week 20 | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| Change from baseline to week 68 | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| PGI-C for Pain | | | | | |
| Week 20 | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| Week 68 | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| PGI-C for PF | | | | | |
| Week 20 | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| Week 68 | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| Body Weight | | | | | |
| Baseline | XX | xx.x (x.xx) | XX.X | xx, xx | xx (xx.x) |
| Week 20 | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| Week 68 | xx | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| Percent change from baseline to week 20 | XX | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |
| Percent change from baseline to week 68 | XX | xx.x (x.xx) | xx.x | xx, xx | xx (xx.x) |

max = maximum; min = minimum; PGI-C = Patient Global Impression of Change; PGI-S = Patient Global Impression of Status; PF = Physical Functioning; SD = standard deviation.

Table A-5. Correlations Between WOMAC Pain, WOMAC Physical Functioning, and SF-36v2 Physical Functioning Scores and Supporting Measures

| | Correlation | Correlation with change in supporting measure, n | |
|---|---|---|---|
| Time/change | PGI-S change | PGI-C | % weight change |
| Change from baseline | to week 20 | | |
| WOMAC Pain | 0.xx*, xx | 0.xx*, xx | 0.xx*, xx |
| WOMAC PF | 0.xx*, xx | 0.xx*, xx | 0.xx*, xx |
| SF-36v2 PF | 0.xx*, xx | 0.xx*, xx | 0.xx*, xx |
| Change from baseline | to week 68 | | |
| WOMAC Pain | 0.xx*, xx | 0.xx*, xx | 0.xx*, xx |
| WOMAC PF | 0.xx*, xx | 0.xx*, xx | 0.xx*, xx |
| SF-36v2 PF | 0.xx*, xx | 0.xx*, xx | 0.xx*, xx |

<sup>\*</sup> P < 0.05 test for H0:  $\rho = 0$ .

PF = Physical Functioning; PGI-C = Patient Global Impression of Change; PGI-S = Patient Global Impression of Status; SF-36v2 = SF-36 Health Survey, Acute Version 2.0; WOMAC = Western Ontario and McMaster Universities Arthritis Index.

Table A-6. Descriptive Statistics of the Changes in WOMAC and SF-36v2 Subscale Scores by Changes in Candidate Anchor Measures

| | Change in WOMAC Pain, WOMAC PF, or SF-36v2 PF | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Time/change/anchor | Mean (SD), n | P10 | P25 | Median | P75 | P90 | Min, max | 95% CI |
| Change from baseline to week 20 | | | | | | | | |
| By change in PGI-S | | | | | | | | |
| < 4-point improvement> | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| 3-point improvement | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| 2-point improvement | xx.x (x.xx), xx | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x, xx.x | xx.x-xx.x |
| 1-point improvement | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| No difference | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| 1-point worsening | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | XX.X-XX.X |
| 2-point worsening | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| 3-point worsening | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | XX.X-XX.X |
| < 4-point worsening> | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| By PGI-C | | | | | | | | |
| Much better | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| Moderately better | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| A little better | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| No difference | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | XX.X-XX.X |
| A little worse | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| Moderately worse | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| Much worse | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | XX.X-XX.) |

| | • | Change | e in WOM/ | AC Pain, W | OMAC PI | F, or SF-3 | 86v2 PF | |
|---|---|---|---|---|---|---|---|---|
| Time/change/anchor | Mean (SD), n | P10 | P25 | Median | P75 | P90 | Min, max | 95% CI |
| By percent change in body weight category (reduction) | | | | | | | | |
| < 5% | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| 5%-10% | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| > 10% | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| Change from baseline to week 68 | l | | | | | | | |
| By change in PGI-S | | | | | | | | |
| < 4-point improvement> | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| 3-point improvement | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| 2-point improvement | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| 1-point improvement | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| No difference | xx.x (xx.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| 1-point worsening | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| 2-point worsening | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| 3-point worsening | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| < 4-point worsening> | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |

| | | Change | e in WOM | AC Pain, W | OMAC PI | F, or SF-3 | 6v2 PF | |
|---|---|---|---|---|---|---|---|---|
| Time/change/anchor | Mean (SD), n | P10 | P25 | Median | P75 | P90 | Min, max | 95% CI |
| By PGI-C | | | | | | | | |
| Much better | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| Moderately better | xx.x (x.xx), xx | xx.x | xx.x | хх.х | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| A little better | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| No difference | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| A little worse | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x-xx.x |
| Moderately worse | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x, xx.x |
| Much worse | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x, xx.x |
| By percent change in body weight category (reduction) | | | | | | | | |
| < 5% | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x, xx.x |
| 5%-10% | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x, xx.x |
| > 10% | xx.x (x.xx), xx | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x, xx.x | xx.x, xx.x |

CI = confidence interval; PF = Physical Functioning; PGI-C = Patient Global Impression of Change; PGI-S = Patient Global Impression of Status; SD = standard deviation; SF-36v2 = SF-36 Health Survey, Acute Version 2.0; WOMAC = Western Ontario and McMaster Universities Arthritis Index.

Notes: This table will be repeated for the changes in WOMAC Pain, WOMAC PF, and SF-36v2 PF subscales and corresponding anchor measures. PGI-S for Pain has up to 3-point changes, while the PGI-S for PF has up to 4-point changes.

Table A-7. Frequencies and Percentages of Crosstabulation Between Changes in PGI-S and PGI-C Items at Week 68

| | • | • | PG | I-C at wee | k 68 | | • |
|---|---|---|---|---|---|---|---|
| Change | Much<br>better | Moderately<br>better | A little<br>better | No<br>difference | a little<br>eworse | Moderately<br>worse | Much<br>worse |
| Change in PGI-S for<br>Pain | | | | | | | |
| 3-point improvement | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 2-point improvement | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 1-point improvement | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| No difference | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 1-point worsening | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 2-point worsening | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 3-point worsening | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Change in PGI-S for<br>PF | | | | | | | |
| 4-point improvement | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 3-point improvement | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 2-point improvement | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 1-point improvement | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| No difference | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 1-point worsening | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 2-point worsening | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 3-point worsening | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| 4-point worsening | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |

PF = Physical Functioning; PGI-C = Patient Global Impression of Change; PGI-S = Patient Global Impression of Status.

Table A-8. Change in WOMAC Pain in Patients Who Achieved a 1-Point PGI-S for Pain Improvement From Baseline to Week 68

| | Baseline PGI-S for Pain | | | |
|---|---|---|---|---|
| Change from baseline to week 68 | Mild | Moderate | Severe | Total |
| n | xx | xx | xx | xx |
| 10th Percentile | xx.x | xx.x | xx.x | xx.x |
| 25th Percentile | xx.x | xx.x | xx.x | xx.x |
| Median | xx.x | xx.x | xx.x | xx.x |
| 75th Percentile | xx.x | xx.x | xx.x | xx.x |
| 90th Percentile | xx.x | xx.x | xx.x | xx.x |

PGI-S = Patient Global Impression of Status; WOMAC = Western Ontario and McMaster Universities Arthritis Index.

Table A-9. Change in WOMAC Pain in Patients Who Achieved a 2-Point PGI-S for Pain Improvement From Baseline to Week 68

| | Baseline PGI-S for Pain | | |
|---|---|---|---|
| Change from baseline to week 68 | Moderate | Severe | Total |
| n | xx | xx | xx |
| 10th Percentile | xx.x | xx.x | xx.x |
| 25th Percentile | xx.x | xx.x | xx.x |
| Median | xx.x | xx.x | xx.x |
| 75th Percentile | xx.x | xx.x | xx.x |
| 90th Percentile | xx.x | xx.x | xx.x |

PGI-S = Patient Global Impression of Status; WOMAC = Western Ontario and McMaster Universities Arthritis Index.

Table A-10. Change in WOMAC and SF-36v2 Physical Functioning in Patients Who Achieved a 1-Point PGI-S for PF Improvement From Baseline to Week 68

| | | Baseline PGI-S for PF | | | |
|---|---|---|---|---|---|
| Change from baseline to week 68 | Poor | Fair | Good | Very<br>good | Total |
| WOMAC PF | | | | | |
| n | XX | xx | xx | xx | xx |
| 10th Percentile | xx.x | xx.x | xx.x | xx.x | xx.x |
| 25th Percentile | xx.x | xx.x | xx.x | xx.x | xx.x |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| 75th Percentile | xx.x | xx.x | xx.x | xx.x | xx.x |
| 90th Percentile | xx.x | xx.x | xx.x | xx.x | xx.x |
| SF-36v2 PF | | | | | |
| n | XX | XX | xx | XX | xx |
| 10th Percentile | xx.x | xx.x | xx.x | xx.x | xx.x |
| 25th Percentile | xx.x | xx.x | xx.x | xx.x | xx.x |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| 75th Percentile | xx.x | xx.x | xx.x | xx.x | xx.x |
| 90th Percentile | xx.x | xx.x | xx.x | xx.x | xx.x |

PF = Physical Functioning; PGI-S = Patient Global Impression of Status; SF-36v2 = SF-36 Health Survey, Acute Version 2.0; WOMAC = Western Ontario and McMaster Universities Arthritis Index.

Table A-11. Change in WOMAC and SF-36v2 Physical Functioning in Patients Who Achieved a 2-Point PGI-S for PF Improvement From Baseline to Week 68

| | Baseline | PGI-S for PF | | |
|---------------------------------|----------|--------------|------|-------|
| Change from baseline to week 68 | Poor | Fair | Good | Total |
| WOMAC PF | | | | |
| n | xx | xx | xx | xx |
| 10th Percentile | xx.x | xx.x | xx.x | xx.x |
| 25th Percentile | xx.x | xx.x | xx.x | xx.x |
| Median | xx.x | xx.x | xx.x | xx.x |
| 75th Percentile | xx.x | xx.x | xx.x | xx.x |
| 90th Percentile | xx.x | xx.x | xx.x | xx.x |
| SF-36v2 PF | | | | |
| n | xx | xx | xx | xx |
| 10th Percentile | xx.x | xx.x | xx.x | xx.x |
| 25th Percentile | xx.x | xx.x | xx.x | xx.x |
| Median | xx.x | xx.x | xx.x | xx.x |
| 75th Percentile | xx.x | xx.x | xx.x | xx.x |
| 90th Percentile | xx.x | xx.x | xx.x | xx.x |

PF = Physical Functioning; PGI-S = Patient Global Impression of Status; SF-36v2 = SF-36 Health Survey, Acute Version 2.0; WOMAC = Western Ontario and McMaster Universities Arthritis Index.

Table A-12. Interpretation of Change: Distribution-Based Method

| Measure | Half-SD at Baseline |
|------------|---------------------|
| WOMAC Pain | x.xx |
| WOMAC PF | x.xx |
| SF-36v2 PF | x.xx |

PF = Physical Functioning; SD = standard deviation; SF-36v2 = SF-36 Health Survey, Acute Version 2.0; WOMAC = Western Ontario and McMaster Universities Arthritis Index.

## **Appendix B. Figure Templates**



Figure B-1. Empirical Cumulative Distribution Function Plot of Change in Target Clinical Outcome Assessment Score, by Change in Anchor Measure

| | • | 10th | 25th | • | 75th | 90th |
|---|---|---|---|---|---|---|
| Change/anchor | n | percentile | percentile | Median | percentile | percentile |
| Change in target COA score | | | | | | |
| Level 1 | XX | xx.x | xx.x | xx.x | xx.x | xx.x |
| Level 2 | XX | xx.x | xx.x | xx.x | xx.x | xx.x |
| Level 3 | xx | xx.x | xx.x | xx.x | xx.x | xx.x |
| Level 4 | XX | xx.x | xx.x | xx.x | xx.x | xx.x |
| | xx | xx.x | xx.x | xx.x | xx.x | xx.x |
| Level k | XX | xx.x | XX.X | xx.x | xx.x | xx.x |

CI = confidence interval; COA = clinical outcome assessment.

Notes: The shaded bands are the 95% CIs of selected change levels of the anchor measure. This figure will be used and repeated only for the change in every target COA score by the changes in appropriate anchor measures from baseline to week 68.



Figure B-2. Probability Density Function Plot of Change in Target Clinical Outcome Assessment Score, by Anchor Measure

 ${\sf CI}$  = confidence interval;  ${\sf COA}$  = clinical outcome assessment.

Notes: The kernel densities are estimated via normal weight functions with the standardized bandwidth = 0.79 x interquartile range x  $\text{n}^{-1/5}$ ; vertical solid lines denote means of different curves as specified in the legend, and vertical dashed lines are the 95% CIs of selected means. This figure will be used and repeated only for the change in every target COA score by the changes in appropriate anchor measures from baseline to week 68.

## 0306398 WOMAC and SF-36 Meaningful Change Final PAP\_24Jan2022

Final Audit Report 2022-02-02 Created: 2022-02-02 Ву: Status: Signed Transaction ID: CBJCHBCAABAAZraO2sTTNSjVAnn0PVneCE-VFmXtxRXP "0306398 WOMAC and SF-36 Meaningful Change Final PAP\_2 4Jan2022" History Document created by 2022-02-02 - 1:47:23 PM GMT Document emailed to for signature 2022-02-02 - 1:49:35 PM GMT Document emailed to for signature 2022-02-02 - 1:49:35 PM GMT Document emailed to for signature 2022-02-02 - 1:49:35 PM GMT Email viewed by 2022-02-02 - 1:52:20 PM GMT Document e-signed by Signature Date: 2022-02-02 - 1:53:23 PM GMT - Time Source: server Email viewed by 2022-02-02 - 2:06:21 PM GMT Document e-signed by Signature Date: 2022-02-02 - 2:06:54 PM GMT - Time Source: server Email viewed by 2022-02-02 - 8:35:03 PM GMT Document e-signed by Signature Date: 2022-02-02 - 8:35:43 PM GMT - Time Source: server 📜 Adobe Sign

